Official Title: A 26-week Randomized, Double-blind, Controlled, Parallel-

group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin compared to Empagliflozin, and Placebo in Patients with Type 2 Diabetes Who Have Inadequate Glycemic Control on Dipeptidyl Peptidase 4 Inhibitor (DPP4(i)) With or Without

Metformin

NCT Number: NCT03351478

**Document Date:** SAP Version 3: 15-November-2019

# Lexicon Pharmaceuticals, Inc.

Sotaglifozin/ LX4211

Protocol No.: EFC14867

A 26-week Randomized, Double-blind, Controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin compared to Empagliflozin, and Placebo in Patients with Type 2 Diabetes Who Have Inadequate Glycemic Control on Dipeptidyl Peptidase 4 Inhibitor (DPP4 (i)) With or Without Metformin

Covance Study ID: 000000155204

**Statistical Analysis Plan** 

Version: 3

DATE OF ISSUE: 15-Nov-2019

Author:

# APPROVALS

The undersigned agree that all required reviews of this document are complete, and approve this Statistical Analysis Plan as final. Programming of the tables, figures and listings based upon the specifications within this document can proceed.

| Covance Amproval: Signature Printed Name/Title | 15 Nov 2019<br>Date |
|---|---|
| Lexicon Approval: | |
| Signature | Date |
| Printed Name/Title | |
| Signature | 15-Nov-7019<br>Date |
| MS, FRS, | # 1 for 12 for the first and a second and a form |
| Signature | SNOV 2019 |
| MD, | Bull to the |
| Printeti Nama | 15-NOV-2019<br>Date |
| Signature | Date |
| PhD, | |
| Printed Name/Title | |

# **TABLE OF CONTENTS**

| LIST OF | F ABBREVIATIONS AND DEFINITION OF TERMS | 6 |
|---|---|---|
| 1 | OVERVIEW AND INVESTIGATIONAL PLAN | 8 |
| 1.1 | STUDY DESIGN AND RANDOMIZATION | 3 |
| 1.2 | OBJECTIVES | 3 |
| 1.2.1 | Primary objectives | 8 |
| 1.2.2 | Secondary objectives | 8 |
| 1.2.3 | Other objectives | S |
| 1.2.4 | Objectives of ABPM substudy | 10 |
| 1.3 | DETERMINATION OF SAMPLE SIZE | 10 |
| 1.4 | STUDY PLAN | 11 |
| 1.5 | MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL | 11 |
| 1.6 | STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN | 12 |
| 2 | STATISTICAL AND ANALYTICAL PROCEDURES | 15 |
| 2.1 | ANALYSIS ENDPOINTS | 15 |
| 2.1.1 | Demographic and baseline characteristics | 15 |
| 2.1.2 | Prior or concomitant medications. | |
| 2.1.2.1 2.1.2.2 | Rescue therapy | |
| 2.1.2.2 | Prohibited prior and concomitant medications | |
| 2.1.3 | Efficacy endpoints Primary efficacy endpoint(s) | |
| 2.1.3.2 | Secondary efficacy endpoint(s) | |
| 2.1.3.3 | Other efficacy endpoint(s) | |
| 2.1.3.4 | ABPM substudy efficacy endpoint(s) | |
| 2.1.4<br>2.1.4.1 | Safety endpoints | |
| 2.1.4.1 | Adverse events variables | |
| 2.1.4.3 | Deaths | |
| 2.1.4.4 | Laboratory safety variables | |
| 2.1.4.5 | Vital signs variables | |
| 2.1.4.6 2.1.4.7 | Physical examination Electrocardiogram variables | |
| 2.1.5 | Pharmacokinetic variables | |
| 2.2 | DISPOSITION OF PATIENTS | 28 |
| 2.2.1 | Randomization and drug dispensing irregularities | 30 |

# Statistical Analysis Plan

| Lexicon F | | Covance Study ID: 000000155204 |
|---|---|---|
| 2.3 | ANALYSIS POPULATIONS | |
| 2.3.1 | Efficacy populations | 31 |
| 2.3.1.1 | Intent-to-treat population | |
| 2.3.1.2 | ABPM substudy population | 32 |
| 2.3.1.3 | Completers population | 32 |
| 2.3.2 | Safety population | 32 |
| 2.3.3 | PK population | 33 |
| 2.4 | STATISTICAL METHODS | 33 |
| 2.4.1 | Demographics and baseline characteristics | 33 |
| 2.4.2 | Prior or concomitant medications | 33 |
| 2.4.3 | Extent of investigational medicinal product exposure and complian | ce34 |
| 2.4.3.1 | Extent of investigational medicinal product exposure | |
| 2.4.3.2 | Compliance | 35 |
| 2.4.4 | Analyses of efficacy endpoints | 36 |
| 2.4.4.1 | Analysis of primary efficacy endpoint | |
| 2.4.4.2 | Analyses of secondary efficacy endpoints | |
| 2.4.4.3 | Analyses of other efficacy endpoints | |
| 2.4.4.4 | Analysis of ABPM substudy efficacy endpoints | |
| 2.4.4.5 | Multiplicity issues | 43 |
| 2.4.5 | Analyses of safety data | 44 |
| 2.4.5.1 | Analyses of hypoglycemia | |
| 2.4.5.2 | Analyses of adverse events | |
| 2.4.5.3 | Deaths | |
| 2.4.5.4 | Analyses of laboratory variables | |
| 2.4.5.5 | Analyses of vital sign variables | |
| 2.4.5.6 | Analyses of electrocardiogram variables | |
| 2.4.5.7 | Analyses of physical examination variables | 52 |
| 2.4.6 | Analyses of pharmacokinetic variables | 52 |
| 2.5 | DATA HANDLING CONVENTIONS | 52 |
| 2.5.1 | General conventions | 52 |
| 2.5.2 | Data handling conventions for secondary efficacy variables | 53 |
| 2.5.3 | Missing data | 53 |
| 2.5.4 | Windows for time points /Measurements for analyses | 56 |
| 2.5.5 | Unscheduled visits | 59 |
| 2.5.6 | Pooling of centers for statistical analyses | 59 |
| 2.5.7 | Statistical technical issues | 59 |
| 3 | INTERIM ANALYSIS | 60 |
| 4 | DATABASE LOCK | 61 |

# Statistical Analysis Plan

Version:3

| Lexicon Pharma | ceuticals, inc. Protocol No. EFC14867 | Covance Study ID: 000000155204 |
|---|---|---|
| 5 SOF | TWARE DOCUMENTATION | 62 |
| 6 REFE | ERENCES | 63 |
| 7 LIST | OF APPENDICES | 64 |
| APPENDIX A | AMBULATORY BLOOD PRESSURE MONITORING SUBS | TUDY65 |
| APPENDIX B | ABPM SUBSTUDY EFFICACY VARIABLE DERIVATION | 68 |
| APPENDIX C | LIST OF PTS FOR SELECT EOSIS (MEDDRA V22.0) | 70 |
| APPENDIX D | POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALIT | IES CRITERIA79 |
| APPENDIX E | SUMMARY OF STATISTICAL ANALYSES | 85 |
| APPENDIX F | STUDY FLOW CHART | 90 |

Date of Issue: 15-Nov-2019

Date of Issue: 15-Nov-2019 Lexicon Pharmaceuticals Protocol No. EFC14867 Covance Study ID: 000000155204

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

ABPM: ambulatory blood pressure monitoring

ACR: albumin-creatinine ratio

AEs: adverse events

adverse events of special interest AESI:

alkaline phosphatase ALP: ALT: alanine aminotransferase ANCOVA: analysis of covariance aspartate aminotransferase AST: ATC: anatomical therapeutic chemical

body mass index BMI: BP: blood pressure BUN: blood urea nitrogen

clinical endpoint committee CEC:

confidence interval CI:

CMH: Cochran-Mantel-Haenszel CPK: creatine phosphokinase clinical study report CSR: CV: cardiovascular

DBP: diastolic blood pressure

DCCT: diabetes control and complications trial

drug-induced liver injury DILI: Data monitoring Committee DMC: DPP4(i): dipeptidyl peptidase 4 inhibitor

electrocardiogram ECG:

e-CRF: electronic case report form

estimated glomerular filtration rate eGFR:

EMA/PRAC: European Medicines Agency/ Pharmacovigilance Risk Assessment Committee

EOSI: events of special interest fasting plasma glucose FPG: glucose-creatinine ratio GCR:

HbA1c: hemoglobin A1c

high density lipoprotein cholesterol HDL-C:

high level group term HLGT: HLT: high level term HR: heart rate

International Federation of Clinical Chemistry and Laboratory Medicine IFCC:

investigational medicinal product IMP: interactive response technology IRT:

intent-to-treat ITT:

#### Statistical Analysis Plan

Version:3

Lexicon Pharmaceuticals Protocol No. EFC14867

Date of Issue: 15-Nov-2019
Covance Study ID: 000000155204

KM: Kaplan-Meier

LDH: lactic acid dehydrogenase

LDL-C: low density lipoprotein cholesterol

LLT: lower level term

MACE: major adverse cardiovascular events

MAR: missing at random

MDRD: modification of diet in renal disease

MedDRA: Medical Dictionary for Regulatory Activities

MI: multiple imputation
MMTT: mixed meal tolerance test
MNAR: missing not at random

NIMP: noninvestigational medicinal product

PCSA: potentially clinically significant abnormality

PPG: postprandial glucose PRA: plasma renin activity

PT: preferred term

SAE: serious adverse events
SAP: statistical analysis plan
SBP: systolic blood pressure
SOC: system organ class
T2D: type 2 diabetes mellitus

TC: total cholesterol

TEAE: treatment-emergent adverse event

TG: triglycerides

UGE: urinary glucose excretion ULN: upper limit of normal

WHO-DD: World Health Organization-Drug Dictionary

# Lexicon Pharmaceuticals Protocol No. EFC14867

#### 1.1 STUDY DESIGN AND RANDOMIZATION

OVERVIEW AND INVESTIGATIONAL PLAN

This is a Phase 3, multicenter and multinational, double blind, placebo- and active-controlled, parallel-group study. Patients will be randomly assigned 2:2:1 to the following 3 treatment groups:

- Sotagliflozin 400 mg.
- Empagliflozin 25 mg.
- Placebo.

The study comprises an up to 4-week Screening Period (consisting of a Screening Phase of up to 2 weeks and a 2-week single-blind placebo Run-in Phase), a 26-week Double-blind Treatment Period, and a 4-week post-treatment Follow-up Period.

At the end of the screening period, eligible patients will be centrally randomized (using permuted block randomization schedule) via an Interactive Response Technology (IRT). The randomization will be stratified by:

- Hemoglobin A1c (HbA1c) at Screening ( $\leq 8.5\%$ , > 8.5%).
- Metformin use at Screening (Yes, No).
- Systolic blood pressure (SBP) at Screening (<130 mmHg, ≥130 mmHg).

It is anticipated to randomize a total of approximately 700 patients. To ensure an approximately equal number of patients have Screening SBP <130 mmHg or SBP ≥130 mmHg, the number of patients enrolled in each category will be limited to 60% of all patients (≤420 patients).

At the preselected study sites participating in the ABPM substudy, approximately 180 of the 700 enrolled patients are expected to participate in an Ambulatory Blood Pressure Monitoring (ABPM) substudy where patients will have blood pressure measured by a validated ABPM device.

#### 1.2 **OBJECTIVES**

## 1.2.1 Primary objectives

The primary objective of this study is to demonstrate the superiority of sotagliflozin 400 mg versus placebo on HbA1c reduction at Week 26 in patients with type 2 diabetes mellitus (T2D) who have inadequate glycemic control on a DPP4(i) with or without metformin.

#### 1.2.2 Secondary objectives

The secondary objectives of this study are to demonstrate:

- Noninferiority of sotagliflozin 400 mg versus empagliflozin on HbA1c reduction from Baseline at Week 26.
- Superiority of sotagliflozin 400 mg versus placebo with respect to:
  - Change from Baseline in 2-hour postprandial glucose (PPG) reduction following a mixed meal tolerance test (MMTT) at Week 26,
  - Change from Baseline in fasting plasma glucose (FPG) reduction at Week 26,
  - Change from Baseline in Body weight reduction at Week 26,
  - Proportion of patients with HbA1c <6.5% and <7.0% at Week 26,
  - Change from baseline in sitting SBP reduction at Week 12 in Patients with SBP≥130 mmHg at Baseline,
  - Change from baseline in sitting SBP reduction at Week 12 in all patients.
- Superiority of sotagliflozin 400 mg versus empagliflozin with respect to change from baseline in:
  - HbA1c reduction at Week 26,
  - Sitting SBP reduction at Week 12 in patients with SBP ≥130 mmHg at Baseline,
  - Sitting SBP reduction at Week 12 in all patients.
- To evaluate the safety of sotagliflozin 400 mg versus empagliflozin 25 mg, and placebo, throughout the 26-week trial.

# 1.2.3 Other objectives

Other objectives of this study are:

- To compare sotagliflozin versus empagliflozin and placebo with respect to change from Baseline in:
  - Estimated glomerular filtration rate (eGFR),
  - Serum creatinine,
  - Urinary glucose excretion (UGE) and urine glucose-creatinine ratio (GCR),
  - Urine albumin-creatinine ratio (ACR) for all patients and patients with urine ACR>30 mg/g at Baseline,
  - Sitting SBP for patients with Baseline SBP <130 mmHg at Weeks 12 and 26,
  - Sitting SBP for patients with Baseline SBP ≥130 mmHg at Week 26,
  - Sitting SBP for all patients at Week 26,
  - Sitting diastolic blood pressure (DBP) for patients with Baseline SBP ≥130 mmHg at Weeks 12 and 26,
  - Reduction in body weight by  $\geq 2\%$ ,  $\geq 5\%$ , and  $\geq 10\%$ .
- To compare sotagliflozin versus empagliflozin with respect to change from Baseline in:

- 2-hour PPG reduction following an MMTT at Week 26,
- FPG reduction at Week 26,
- Body weight reduction at Week 26.
- To compare the use of rescue medications for hyperglycemia in the sotagliflozin and empagliflozin treatment groups.
- To assess plasma levels of sotagliflozin and sotagliflozin-3-O-glucuronide in the sotagliflozin treatment arm.
- To compare hemodynamic markers (including plasma renin activity (PRA), aldosterone, angiotensinogen 1, angiotensinogen 2 and glucagon) in the sotagliflozin and empagliflozin treatment groups.

# 1.2.4 Objectives of ABPM substudy

The objective of the ABPM substudy is to compare the effect of sotagliflozin, empagliflozin and placebo in a subset of patients based on:

- 24-hour average SBP and DBP.
- Average adjusted awake time blood pressure (BP) as measured by SBP and DBP with adjustment based on actigraphy.
- Average adjusted sleeping time BP as measured by SBP and DBP with adjustment based on actigraphy.

Full details of the ABPM substudy are provided in Appendix A.

#### 1.3 DETERMINATION OF SAMPLE SIZE

The sample size/power calculations were performed based on the primary endpoint.

A sample size of 280 patients in the sotagliflozin group and 140 patients in the placebo group will provide more than 90% power to detect a difference of 0.6% for change from Baseline to Week 26 in HbA1c between sotagliflozin and placebo (standard deviation [SD]=1.1%; 5% significance level 2-sided).

A sample size of 280 patients in the sotagliflozin group and 280 patients in the empagliflozin group will ensure that the upper bound of the 2-sided 95% CI of the adjusted mean difference would not exceed 0.3% with more than 80% power to show noninferiority for intent-to-treat (ITT) analysis and for completer analysis considering 15% dropout. This calculation assumes a common SD of 1.1%, and the true difference between sotagliflozin and empagliflozin is zero for change from Baseline to Week 26 in HbA1c.

The total sample size will be approximately 700 patients to be randomized (sotagliflozin group: 280; empagliflozin group: 280; placebo group: 140).

#### 1.4 STUDY PLAN

The study plan is presented graphically as follows.



The study flowchart can be found in Appendix F.

## 1.5 MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL

This section summarizes major changes to the protocol statistical section with emphasis on changes after study start (after the first patient was enrolled).

The protocol history table below gives the timing, rationale, and key details of major changes to the protocol statistical section.

The first patient was enrolled on 27-Nov-2017. There were no planned interim analyses.

Table 1 - Protocol amendment statistical changes

| Amendment<br>Number | Date<br>Approved | Rationale | Description of statistical changes |
|---|---|---|---|
| 2 | 11-April-2018 | The actigraphy capacity of the ABPM device will be used to measure the patient's activity levels, ie, when he/she is awake or asleep. This will provide a more accurate assessment of awake time and sleeping time BP, because not all patients have the same activity/sleeping patterns. | Objectives and endpoints of ABPM substudy updated: Average adjusted awake time BP and sleeping time BP modified as measured by SBP and DBP with adjustment based on actigraphy |
| 2 | 11-April-2018 | Baseline eGFR defined as<br>recommended by CDISC<br>Therapeutic Area Data Standards<br>User Guide for Diabetic Kidney<br>Disease | For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP for those randomized and exposed or before randomization for those who were randomized but never exposed to IMP. |
| 2 | 11-April-2018 | For some sites the standard meal supplies are not approved by the local regulatory agency, the patients will not participate in the MMTT. | Those patients in the sites of specific region will not be included in the efficacy population for MMTT analyses. No such specific region exists, so this amendment does not change the statistical analysis. See Section 1.6. |

## 1.6 STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN

The statistical analysis plan (SAP) history table below gives the timing, rationale, and key details for major changes to the statistical analysis features in the statistical analysis plan. Changes also incorporated in a protocol amendment are cross-referenced to Table 1.

Table 2 - Statistical analysis plan statistical changes

| Table 2 - Statistical analysis plan statistical changes | | | |
|---|---|---|---|
| SAP<br>version<br>number | Date<br>approved | Rationale | Description of statistical changes |
| 1 | 04-Oct-2018 | The actigraphy capacity of the ABPM device will be used to measure the patient's activity levels, ie, when he/she is awake or asleep. This will provide a more accurate assessment of awake time and sleeping time BP, because not all patients have the same activity/sleeping patterns. | Objectives and endpoints of ABPM substudy updated: Average adjusted awake time BP and sleeping time BP modified as measured by SBP and DBP with adjustment based on actigraphy* |
| 1 | 04-Oct-2018 | Baseline eGFR defined as recommended by CDISC Therapeutic Area Data Standards User Guide for Diabetic Kidney Disease | For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP for those randomized and exposed or before randomization for those who were randomized but never exposed to IMP* |
| 1 | 04-Oct-2018 | Clarification on EOSI renal events | Details specified on renal events to be consistent with outcome studies in Section 2.1.4.2. |
| 1 | 04-Oct-2018 | | |
| 1 | 04-Oct-2018 | | |
| 1 | 04-Oct-2018 | No such sites that the standard meal supplies are not approved by the local regulatory agency. | Remove the statement that those patients in the specific region will not be included in the efficacy population for MMTT analyses. Efficacy population will be used for MMTT analyses |
| 1 | 04-Oct-2018 | Updating the wording to be consistency with CEC charter | Unstable angina leading to hospitalization changed to Unstable angina requiring hospitalization |
| 2 | 11-Jun-2019 | | |
| 2 | 11-Jun-2019 | Number of iterations for multiple imputation was changed | Number of iterations for multiple imputation was changed from 10 000 to 2000 |
| 2 | 11-Jun-2019 | Wording change to be consistent with CEC charter | "Heart failure leading to hospitalization" changed to "Heart failure requiring hospitalization" |
| 2 | 11-Jun-2019 | MedDRA version and dictionary updated | MedDRA version was updated to V22.0 and list of PTs for selected EOSI was updated |
| 2 | 11-Jun-2019 | To add high and low doses of vildagliptin for baseline characteristics | Label recommended high and low doses added for vildagliptin |

| SAP | | | |
|---|---|---|---|
| version | Date | | |
| number | approved | Rationale | Description of statistical changes |
| 3 | This version | | |
| 3 | This version | | |
| 3 | This version | | |
| 3 | This version | | |
| 3 | This version | Assess robustness on the ITT-based analyses | Identify possible need to conduct sensitivity<br>analyses for PK anomalies |
| 3 | This version | Compare treatment groups for<br>important pharmacodynamic<br>measures | Addition of inferential analyses for UGE and UGCR endpoints |
| 3 | This version | Maximize number of null hypotheses to reject, include/omit clinically meaningful hypotheses to test | Analyses of some secondary endpoints are omitted from the statistical testing hierarchy: FPG reduction at week 26 (superiority comparison of sotaglifozin 400 versus placebo), |
| | | | HbA1c responder analysis (HbA1c < 7.0% at Week 26 / superiority comparison of sotaglifozin 400 versus placebo), |
| | | | Sitting SBP reduction at Week 12 (superiority comparison of sotaglifozin 400 versus placebo) |
| | | | Addition of 2-Hour PPG reduction at Week 26 as a secondary endpoint to statistical testing hierarchy (superiority comparison of sotagliflozin 400 mg versus empagliflozin 25 mg) |

<sup>\*</sup> Change made in Protocol Amendment 2 dated 11-April-2018.

# 2 STATISTICAL AND ANALYTICAL PROCEDURES

#### 2.1 ANALYSIS ENDPOINTS

#### 2.1.1 Demographic and baseline characteristics

The baseline value (with the exception of serum creatinine and eGFR) is defined as the last available value before the first dose of double-blind investigational medicinal product (IMP), or the last available value prior to randomization for patients who were randomized but never exposed to IMP.

For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP for those randomized and exposed or before randomization for those who were randomized but never exposed to IMP.

Baseline safety and efficacy parameters are presented along with the summary statistics in the safety and efficacy sections (Section 2.4.5 and Section 2.4.4).

#### Demographic characteristics

Demographic characteristics to be summarized are:

- Age (years) derived as: (Year of informed consent Year of birth).
- Age categories:  $(<50, \ge 50 \text{ to } <65, \ge 65 \text{ to } <75, \ge 75 \text{ years})$ .
- Gender (Male, Female).
- Race (White, Black or African American, Asian, American Indian or Alaska native, Native Hawaiian or other pacific islander, Multiple, Unknown).
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Unknown).
- HbA1c (%) at screening visit.
- Randomization strata of HbA1c ( $\leq 8.5\%$ , > 8.5%) at screening (data from IRT).
- Randomization strata of metformin use (Yes, No) at screening (data from IRT).
- Mean SBP at screening.
- Randomization strata of SBP (<130 mmHg, ≥130 mmHg) at screening (data from IRT).
- Baseline body mass index (BMI) (kg/m<sup>2</sup>) derived as: (Weight in kg)/(Height in meters)<sup>2</sup>.
- Baseline BMI categories ( $<30, \ge 30 \text{ kg/m}^2$ ).
- Country.

# Disease characteristics at screening or baseline

# Disease history includes:

- Duration of diabetes (years) derived as: (Date of informed consent Date of diagnosis of diabetes + 1)/365.25.
- Duration of diabetes categories:  $(<10, \ge 10 \text{ years})$ .
- Age at diagnosis of diabetes (years): (Year of diagnosis of diabetes Year of birth).
- Metformin use at screening (Yes, No).
- Duration of metformin treatment (for those patients who used metformin at screening) (years): (date of informed consent date of first intake of metformin +1)/365.25.
- Daily dose of metformin (mg) at baseline (for those patients who used metformin at screening).
- Categorized daily dose of metformin at baseline for those patients who used metformin at screening (<1500,  $\ge 1500$  to <2500,  $\ge 2500$  mg).
- Duration of DPP4(i) treatment (years): (date of informed consent date of first intake of DPP4(i) +1)/365.25.
- Categorized daily dose of DPP4(i) at baseline:
  - At label recommended high dose,
  - At label recommended low dose,
  - Other doses.

where the label recommended high dose for sitagliptin is 100 mg, alogliptin is 25 mg, saxagliptin is 5 mg, linagliptin is 5 mg and vildagliptin is 100 mg, and label recommended low dose for sitagliptin is 50/25 mg, alogliptin is 12.5 mg, saxagliptin is 2.5 mg and vildagliptin is 50 mg.

- Baseline diabetic microvascular complications (Yes, No) [ie, diabetic retinopathy, diabetic neuropathy, diabetic peripheral neuropathy (sensory or motor), diabetic autonomic neuropathy, diabetic foot infection].
- Baseline urine ACR categories (<30 mg/g [Normal], ≥30 to <300 mg/g [Microalbuminuria], and ≥300 mg/g [Macroalbuminuria]).
- eGFR at screening (mL/min/1.73m<sup>2</sup>).
- eGFR categories at screening (<15 mL/min/1.73m² [End stage renal disease], ≥15 to <30 mL/min/1.73m² [Severe decrease in GFR], ≥30 to <60 mL/min/1.73m² [Moderate decrease in GFR], ≥60 to <90 mL/min/1.73m² [Mild decrease in GFR], and ≥90 mL/min/1.73m² [Normal]).
- Prior antihypertensive medication identified by therapeutic class as agents acting on the renin-angiotensin system, beta blocking agents, diuretics (a sub-category: loop diuretics identified by pharmacological class as high-ceiling diuretics), calcium channel blockers,

and antihypertensives according to World Health Organization-Drug Dictionary (WHO-DD).

## Medical or surgical history

Medical history and medical findings include:

- Physical examination.
- Medical or surgical history.
- Medical history cardiovascular.
- Surgical history amputation.
- Alcohol habits.
- Tobacco smoking habits.

Medical and surgical history will be coded to a "lower level term (LLT)", "preferred term (PT)", "high level term (HLT)", "high level group term (HLGT)", and associated primary "system organ class (SOC)" using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at Covance at the time of database lock.

Any technical details related to computation, dates, and imputations for missing dates are described in Section 2.5.

#### 2.1.2 Prior or concomitant medications

All medications taken within 3 months before the screening visit (any time for prior SGLT2) and until the end of the study are to be reported in the electronic case report form (e-CRF).

All medications will be coded using the WHO-DD using the version currently in effect at Covance at the time of database lock.

- Prior medications are those the patient used prior to first administration of the double-blind IMP. Prior medications can be discontinued before first administration or can be ongoing during treatment phase.
- Concomitant medications are any treatments received by the patient concomitantly to any IMP, from first administration of double-blind IMP to the date of last administration + 10 days. A given medication can be classified both as a prior medication and as a concomitant medication.
- Posttreatment medications are those the patient took in the period running from the 11<sup>th</sup> day after the last administration of double-blind IMP up to the end of the study.

Background DPP4(i) and metformin are considered as noninvestigational medicinal products (NIMP).

Any technical details related to computation, dates, imputation for missing dates are described in Section 2.5.

#### 2.1.2.1 Rescue therapy

If rescue thresholds are reached, Sulfonylurea (eg, glimepiride) should be added first, unless there is a contraindication to sulfonylurea treatment per label. In case of contraindication to sulfonylurea, another rescue medication (oral or injectable) can be added at the Investigator's decision except for SGLT2 inhibitors. Rescue therapy is considered a NIMP.

#### 2.1.2.2 Prohibited prior and concomitant medications

During the study treatment period, the following medications are prohibited:

- Initiation of any antidiabetic agents, including oral or injectable antihyperglycemic agents other than the IMP is not allowed before the rescue therapy. The existing background medication (NIMP) should not be modified before the rescue.
  - **Note:** Short term use (<10 consecutive days) of the prohibited medication, eg, short-acting insulin for treatment of acute illness or surgery, is allowed.
- Systemic use of glucocorticoids is not allowed for more than 10 consecutive days within 90 days prior to the Screening Visit.
  - **Note:** Topical, ophthalmic, nasal spray, or inhaled applications are allowed.
- SGLT2 inhibitors (eg, canagliflozin, dapagliflozin) are not allowed for rescue or post-IMP treatment until the planned end of the study (Visit 9, Week 30).
- Modification of antihypertensive medication before Week 12 is not allowed unless for safety reasons.
- Use of investigational medication in any other clinical study.
- Initiation of any weight loss drugs (eg, phentermine, orlistat).
- Patients taking sotagliflozin with concomitant digoxin should have digoxin concentrations
  monitored and doses reduced as needed. In addition, other P-gp substrates may be affected
  and the labels of P-gp substrate drugs should be consulted with regards to monitoring and
  dose adjustments.

Other medications which are unlikely to interfere with the PKs or pharmacodynamics of the IMP or confound interpretation of the study endpoints are allowed as needed, following discussion between the Investigator and the Sponsor/CRO. However, doses of chronically administered medicines should be kept fixed during the trial if at all possible.

The dose of all antihypertensive agents should be kept constant during the 12 weeks following randomization and no antihypertensive agents should be added or withdrawn for the 12 weeks following randomization unless it is considered necessary for safety reasons.

#### 2.1.3 Efficacy endpoints

All efficacy measurements collected during the study will be considered for analyses, including those obtained after IMP discontinuation or introduction of rescue therapy (see Section 2.5.4).

HbA1c, 2-hour PPG, FPG, urine ACR, UGE, urine GCR, serum creatinine, eGFR and hemodynamic markers are measured/calculated in a central laboratory (see study flowchart in Appendix F). Body weight, SBP and DBP (see Section 2.1.4.4) are measured at on-site visits by the investigator. Patients requiring rescue are identified as those with the reason for treatment ticked "rescue therapy" in e-CRF "Medication" page.

Efficacy variables will be summarized in both standard international units and conventional units when applicable.

# 2.1.3.1 Primary efficacy endpoint(s)

The primary efficacy endpoint is the change from Baseline to Week 26 in HbA1c (%).

## 2.1.3.2 Secondary efficacy endpoint(s)

The secondary efficacy endpoints are:

- Change from Baseline to Week 26 in 2-hour PPG following an MMTT.
- Change from Baseline to Week 26 in FPG.
- Change from Baseline to Week 26 in body weight.
- Proportion of patients with HbA1c <6.5%, <7.0% at Week 26 (HbA1c responders).
- Change from Baseline to Week 12 in sitting SBP in patients with SBP ≥130 mmHg at Baseline.
- Change from Baseline to Week 12 in sitting SBP in all patients.

#### 2.1.3.3 Other efficacy endpoint(s)

Other efficacy endpoints include:

- Change from Baseline in:
  - eGFR.
  - Serum creatinine,
  - UGE and urine GCR,
  - Urine ACR for all patients and patients with Urine ACR >30 mg/g,
  - Sitting SBP for patients with Baseline SBP <130 mmHg at Weeks 12 and 26,
  - Sitting SBP for patients with Baseline SBP ≥130 mmHg at Week 26,
  - Sitting SBP for all patients at Week 26,

- Sitting DBP for patients with Baseline SBP ≥130 mmHg at Weeks 12 and 26,
- Reduction in body weight  $\geq 2\%$ ,  $\geq 5\%$ , and  $\geq 10\%$ .
- Use of rescue medications for hyperglycemia in the sotagliflozin and empagliflozin treatment groups.
- Plasma concentration of sotagliflozin and sotagliflozin-3-O-glucuronide for patients receiving sotagliflozin.
- Hemodynamic markers (including PRA, aldosterone, angiotensinogen 1, angiotensinogen 2 and glucagon).

# 2.1.3.4 ABPM substudy efficacy endpoint(s)

The ABPM endpoints are changes from Baseline to Week 12 and Week 26 for all patients participating substudy, patients with baseline 24-hour average SBP≥130 mmHg and patients with baseline 24-hour average SBP<130 mmHg in:

- 24-hour average SBP and DBP.
- Average adjusted awake time BP as measured by SBP and DBP with adjustment based on actigraphy.
- Average adjusted sleeping time BP as measured by SBP and DBP with adjustment based on actigraphy.

# 2.1.4 Safety endpoints

The safety analysis will be based on the reported adverse events (AEs), hypoglycemia, and other safety information, such as clinical laboratory data, vital signs, electrocardiogram (ECG), and physical examination, etc.

#### Observation period

The observation period will be divided into 4 epochs:

- The **screening** epoch is defined as the time from the signed informed consent date up to the first administration of the double-blind IMP.
- The **treatment** epoch is defined as the time from the first administration of the double-blind IMP to the last administration of the double-blind IMP.
- The **residual treatment** epoch is defined as the time from the last administration of the double-blind IMP up to 10 days (1 day for hypoglycemia) after the last administration of the double-blind IMP.

The treatment-emergent adverse event (TEAE) period will include both **treatment** and **residual treatment** epochs.

• The **posttreatment** epoch is defined as the period of time starting the day after the end of the treatment-emergent adverse event period up to the last protocol-planned visit or the resolution/stabilization of all serious adverse events (SAE), adverse events of special interest (AESI) and events of special interest (EOSI), whichever is later.

The on-study observation period is defined as the time from start of double-blind treatment until the end of the study (defined as the last scheduled visit for those who completed the study and the date collected on e-CRF page "Completion of End of Study/Follow-up" for those who did not complete the study).

The post-study observation period is defined as the time from the day after the end of the study until the resolution/stabilization of all SAE, AESI and EOSI if applicable.

# 2.1.4.1 Hypoglycemia

Hypoglycemia will be identified as events recorded on the dedicated e-CRF "Hypoglycemic event information" page, and will be categorized as follows (see study protocol for further details):

# Severe hypoglycemia

Severe hypoglycemia is an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure, unconsciousness or coma.

Self-monitored plasma glucose values may not be available, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.

Severe hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- 1. To the question "Countermeasure Administration", ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and
- 2. To the question "Were Symptoms Present", ticked "Yes".

## Documented symptomatic hypoglycemia

Documented symptomatic hypoglycemia is an event during which typical symptoms of hypoglycemia accompanied by a measured plasma glucose concentration of  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL).

Clinical symptoms that are considered to result from a hypoglycemic episode are eg, increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, or coma.

Documented symptomatic hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and
- 2. To the question "Were Symptoms Present", ticked "Yes", and
- 3. With a plasma glucose value before countermeasure  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL).

# Asymptomatic hypoglycemia

Asymptomatic hypoglycemia is an event not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose concentration  $\leq$  3.9 mmol/L ( $\leq$ 70 mg/dL).

Asymptomatic hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as.

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and
- 2. To the question "Were Symptoms Present", ticked "No", and
- 3. With a plasma glucose value before countermeasure  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL).

# Probable symptomatic hypoglycemia

Probable symptomatic hypoglycemia is an event during which symptoms of hypoglycemia are not accompanied by a plasma glucose determination, (but that was presumably caused by a plasma glucose concentration  $\leq$ 3.9 mmol/L [ $\leq$ 70 mg/dL]), ie, symptoms treated with oral carbohydrate without a test of plasma glucose.

Probable symptomatic hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and
- 2. To the question "Were Symptoms Present", ticked "Yes", and
- 3. With no plasma glucose value before countermeasure, and
- 4. To the question "Did this countermeasure lead a significant improvement or prompt recovery?", ticked "Yes".

## Relative hypoglycemia

Relative hypoglycemia, recently termed "pseudo-hypoglycemia" is an event during which the patient reports typical symptoms of hypoglycemia, and interprets the symptoms as indicative of hypoglycemia, but with a measured plasma glucose concentration >3.9 mmol/L (>70 mg/dL).

Relative hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance",
- 2. To the question "Were Symptoms Present", ticked "Yes", and
- 3. With a plasma glucose value before countermeasure >3.9 mmol/L (>70 mg/dL).

In addition of the threshold of  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL), hypoglycemia episodes with a plasma glucose of  $\leq$ 3.0 mmol/L ( $\leq$ 54 mg/dL) will be analyzed separately.

Any hypoglycemic event fulfilling the criteria of a SAE or leading to unconsciousness, coma, or seizure will also be recorded as a SAE (see Section 2.1.4.1).

#### 2.1.4.2 Adverse events variables

#### Adverse event observation period

- Pretreatment adverse events are adverse events that developed or worsened or became serious from the signed informed consent date up to first administration of double-blind IMP.
- Treatment-emergent adverse events are adverse events that developed or worsened or became serious during the treatment-emergent adverse event period.
- Posttreatment adverse events are adverse events that developed or worsened or became serious during the posttreatment period.

All adverse events (including SAE, AESI and EOSI) will be coded to a lower-level term (LLT), preferred term (PT), high-level term (HLT), high-level group term (HLGT), and associated primary system organ class (SOC) using the version of MedDRA currently in effect at Covance at the time of database lock.

The occurrence of adverse events (including SAE, AESI and EOSI) will be recorded from the time of signed informed consent until the end of the study (see Section 2.1.4) or the resolution/stabilization of all SAE, AESI and EOSI.

## **AESI** include:

- Pregnancy.
- Symptomatic overdose with IMP/NIMP.
- Alanine aminotransferase (ALT) increase >3 × upper limit of normal (ULN).

#### **EOSI** include:

- Major adverse cardiovascular events (MACE [cardiovascular death, myocardial infarction, or stroke]) and other specific cardiovascular (CV) events (eg, heart failure requiring hospitalization).
- Severe hypoglycemia.

- Genital mycotic infections (to include vulvovaginal candidiasis in females and candida balanitis in males).
- Urinary tract infection.
- Clinically relevant volume depletion and events related/possibly related to volume depletion.
- Diarrhea.
- Pancreatitis.
- Bone fractures.
- Venous thrombotic events, to include deep venous thrombosis and thromboembolism (to include pulmonary embolism).
- Diabetic ketoacidosis.
- Renal events, to include 50% decline in eGFR, end stage kidney disease, renal death.
- Malignancies of special interest (breast, bladder, renal cell, Leydig cell, pancreatic, prostate, and thyroid cancer).
- Adverse event leading to an amputation.

A Clinical Endpoint Committee (CEC) will, in a blinded manner, review and adjudicate all deaths, myocardial infarction, stroke, unstable angina requiring hospitalization, and heart failure requiring hospitalization, selected renal events, bone fracture, and diabetic ketoacidosis.

Two independent committees will review safety events that require ongoing monitoring to ensure timing protocol amendments in case a safety signal is identified. These events are: 1) potential cases of drug-induced liver injury (DILI), and 2) cases of amputations. The two committees will review the cases in a treatment-blinded manner and will present their assessment to the DMC.

AESI and EOSI will be identified based on criteria in Table 3.

Table 3 - Criteria for AESI and EOSI

| AE Grouping | Criteria |
|---|---|
| AESI | |
| Pregnancy | e-CRF "Pregnancy" |
| Symptomatic overdose with IMP/NIMP | "Overdose of IMP" or "Overdose of NIMP" checked and "Symptomatic overdose" checked in e-CRF "Overdose" |
| ALT increase >3 × ULN | e-CRF "ALT increase" |
| EOSI adjudicated | |
| Cardiovascular death | Positively adjudicated by CEC: "Cardiovascular" or "Undetermined" as the primary cause of death |
| Myocardial infarction, Unstable<br>Angina requiring hospitalization | Positively adjudicated by CEC: Yes to the question "Does the event meet the definition of an MI for this study?", or Yes to the question "If event is not an MI, does the event meet the definition of an UA Requiring admission to hospital or emergency room, for this study?" |


| AE Grouping | Criteria |
|---|---|
| Stroke | Positively adjudicated by CEC: Yes to the question "Does the event meet the definition of a Stroke for this study?" |
| Heart failure requiring hospitalization | Positively adjudicated by CEC: Yes to the question "Does the event meet the definition of a Heart Failure Event for this study?" |
| Bone fractures | Positively adjudicated by CEC: Yes to the question "Did the Fracture occur?" |
| Diabetic ketoacidosis | Positively adjudicated by CEC: Yes to the question "Does this event meet the criteria to be a DKA event?" |
| EOSI Renal events where select e | vents adjudicated |
| Sustained ≥50% decrease in | (1) For ≥50% decrease in eGFR from baseline, |
| eGFR | (1a) confirmed ≥50% decrease in GFR for ≥30 days with no reversible cause as recorded in e-CRF "eGFR decrease", OR |
| | (1b) positively adjudicated by CEC: Yes to the question "Does the subject meet the criteria of CKD progression" for ≥50% decrease in eGFR. |
| Sustained eGFR <15 | (2) For eGFR <15 mL/min/1.73 m <sup>2</sup> , |
| mL/min/1.73 m² | (2a) confirmed eGFR <15 mL/min/1.73 m2 for ≥30 days with no reversible cause as recorded in e-CRF "eGFR decrease", OR |
| | (2b) positively adjudicated by CEC: Yes to the question "Does the subject meet the criteria of CKD progression". |
| Chronic dialysis | (3) For dialysis, |
| | (3a) dialysis lasted for ≥90 days (eg, end date – start date+ 1 ≥90) as recorded in e-CRF "Renal Event – Dialysis", OR |
| | (3b) positively adjudicated by CEC: Yes to the question ". Does the subject meet the criteria for ESRD". |
| Renal transplant* | (4) "Renal transplant" captured in e-CRF "Other procedure form", where adjudication is not required. PTs of Renal transplant (10038533), Renal and pancreas transplant (10052278), Renal and liver transplant (10052279) based on MedDRAv22.0. |
| Renal death | (5) Renal death as positively adjudicated by CEC: "Death - Non-Cardiovascular (Renal)" as the primary cause of death |
| EOSI not adjudicated* | |
| Severe hypoglycemia | Algorithm specified in Section 2.1.4.1 based on e-CRF "Hypoglycemic Events" |
| Genital mycotic infections | PTs in Appendix C |
| Urinary tract infections | PTs in Appendix C |
| Clinically relevant volume depletion and events related/possibly related to volume depletion | PTs in Appendix C |
| Diarrhea | Narrow search on "Noninfectious diarrhoea (SMQ)" [20000218] plus the following PTs (MedDRA v22.0: Gastroenteritis (10017888), Antidiarrhoeal supportive care (10055660), Enteritis (10014866), Enteritis leukopenic (10014877), Enterocolitis (10014893), Enterocolitis haemorrhagic (10014896) |
| Pancreatitis | PTs in Appendix C |

| Lexicon Pharmaceuticals Protocol No. EFC14867 | | Covance Study ID: 000000155204 |
|---|---|---|
| AE Grouping | Criteria | |
| Venous thrombotic events | PTs in Appendix C | |
| Malignancies of special interest | Breast cancer: Narrow search on "Breast ne [20000149] | eoplasms, malignant and unspecified (SMQ)" |
| | Prostate cancer: Narrow search on "Prostat [20000152] | te neoplasms, malignant and unspecified (SMQ)" |
| | Leydig-cell cancer: PTs of Leydig cell tumor<br>Sertoli-Leydig cell tumour (10073270) base | , |
| | Thyroid cancer: PTs in Appendix C | |
| | Renal cell cancer: PTs in Appendix C | |
| | Pancreatic cancer: PTs in Appendix C | |
| | Bladder cancer: PTs in Appendix C | |
| EOSI AE leading to an amputati | on | |
| AE leading to an amputation | "AE Correction" as the reason for amputation in e-CRF "Other Procedures related to Amputation" | |
| AE potentially leading to an amputation ** | PTs in Appendix C | |

<sup>\*</sup> Search terms will be updated using the MedDRA version currently in effect at Covance at the time of database lock for EOSI identified by

#### 2.1.4.3 Deaths

The deaths observation period are per the observation periods defined above.

- Death on-study: deaths occurring during the on-study observation period.
- Death on-treatment: deaths occurring during the TEAE period.
- Death post-study: deaths occurring after the end of the study.

## 2.1.4.4 Laboratory safety variables

Clinical laboratory data consists of blood analysis (including hematology, clinical chemistry, amylase, lipase and lipid profile) and urinalysis. Clinical laboratory values will be summarized in both standard international units and conventional units when applicable.

Blood samples for clinical laboratories will be collected at designated visits (see study flowchart in Appendix F). The following laboratory data will be measured at a central laboratory:

- Hematology:
  - Red blood cells and platelets: hemoglobin, hematocrit, red blood cell, platelets count,
  - White blood cells: white blood cell, neutrophils, lymphocytes, monocytes, basophils, eosinophils.

Date of Issue: 15-Nov-2019

<sup>\*\*</sup> AE potentially leading to amputation: not one of EOSI defined in protocol, included and analyzed due to their relevance in regards to lower limb complications and amputations as a requirement from health authorities.

- Clinical chemistry:
  - **Metabolism:** glucose (serum), creatine phosphokinase (CPK),
  - **Electrolytes and minerals**: sodium, potassium, chloride, bicarbonate (ie, carbon dioxide), calcium, phosphorus, magnesium,
  - Renal function: blood urea nitrogen (BUN), creatinine, uric acid,
  - **Liver function**: total protein, albumin, ALT, aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin, Lactic acid dehydrogenase (LDH).
- Lipid parameters (fasting): total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C) (calculated by Friedwald equation, See Section 2.5.1), Non-HDL-C (calculated as the difference between TC and HDL-C), triglycerides (TG).
- Pancreatic enzymes: lipase, amylase.

Urine samples will be collected at designated visits (see study flowchart in Appendix F). The following laboratory data will be measured at a central laboratory:

- Urine dipstick includes: specific gravity, pH, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase
- Urine microscopy includes, but is not limited to: detection of formed cellular elements, casts, bacteria, yeast, parasites, and crystals in centrifuged urine sediment
- Urine albumin, total protein, calcium, glucose, creatinine, phosphorus, and magnesium

Serum glucose, UGE, calculated urine ACR and calculated urine GCR will be presented as efficacy parameters in Section 2.4.4. For creatinine and calculated eGFR, PCSA summaries will be presented in the safety section while descriptive summaries in the efficacy section.

Technical formulas are described in Section 2.5.1.

# 2.1.4.5 Vital signs variables

Vital signs include: heart rate (HR), systolic and diastolic blood pressure, temperature, and respiratory rate (see study flowchart in Appendix F for designated visits). They will be performed after the patient has been seated for at least 5 minutes. Blood pressure and HR will be assessed 3 times with at least 1 minute between each measurement following the 5-minute rest period, and prior to phlebotomy. The mean of the 3 measurements will be analyzed for each vital sign variable (HR, SBP, and DBP).

#### 2.1.4.6 Physical examination

A complete physical exam will be performed at Visit 1 (Screening) and Visit 8 (Week 26). "Normal", "Abnormal" or "Not done" as determined by the Investigator will be reported in the e-CRF by body system.

#### 2.1.4.7 Electrocardiogram variables

12-lead ECGs will be performed at Visit 2 (Run-in) and Visit 8 (Week 26). ECG status of "normal" or "abnormal" will be reported in the e-CRF as determined by the Investigator.

#### 2.1.5 Pharmacokinetic variables

Pharmacokinetic variables include the plasma concentration of sotagliflozin and its 3-O-glucuronide metabolite in the sotagliflozin group.

#### 2.2 DISPOSITION OF PATIENTS

This section describes patient disposition for both patient study status and the patient analysis populations.

Screened patients are defined as all patients who have signed the informed consent.

Randomized patients consist of all patients with a signed informed consent form who have had a treatment kit number allocated and recorded in the IRT database, regardless of whether the treatment kit was used or not.

For patient study status, the total number of patients in each of the following categories will be presented in the clinical study report (CSR) using a flowchart diagram or summary tables:

- Screened patients.
- Run in patients: patients who had a run-in record in IRT.
- Screen failure patients (including failures during run-in) and reasons for screen failure.
- Nonrandomized but treated patients.
- Randomized patients.
- Randomized but not treated patients.
- Randomized and treated patients.
- Patients who have completed the 26-week double-blind treatment period as scheduled.
- Patients who did not complete the 26-week double-blind treatment period as scheduled and the reasons for permanent treatment discontinuation.

- Patients who have completed the study as scheduled.
- Patients who did not complete the study as scheduled and the reasons for study discontinuation.
- Patients' end of study status (completed, not completed) and corresponding end of treatment status (completed, not completed).
- Status at last study contact.

For screened, run in, screen failure, and nonrandomized but treated patients, percentages will be calculated using the number of screened patients as the denominator. All other categories of patients will be presented by treatment group and the percentages will be calculated using the number of randomized patients within each treatment group as the denominator. Reasons for treatment discontinuation will be supplied in tables giving numbers and percentages by treatment group. Patients prematurely discontinued from treatment and/or study, along with reasons for discontinuation, will also be listed.

A summary of the distribution of patients by country and center will also be provided (overall number of patients screened, run-in, randomized, and treated, as well as number of patients randomized, discontinued from study treatment, and discontinued from study for each treatment group).

Patients treated but not randomized, patients randomized but not treated and patients randomized but not treated as randomized will be identified and described in separate listings. The patients of the third category (randomized and not treated as randomized) will be part of efficacy and safety analyses (see Section 2.3). Patients randomized but not treated will be included in efficacy analysis. Safety data of patients treated but not randomized will be reported separately.

The randomization strata [HbA1c at Screening ( $\leq$ 8.5%, >8.5%), metformin use at Screening (Yes, No) and mean SBP at Screening (<130,  $\geq$ 130 mmHg)] assigned by IRT will be summarized. The percentages will be calculated using the number of randomized patients as the denominator. The discrepancy between the strata assigned by IRT and the information reported on e-CRF will be listed for all randomized patients.

Kaplan-Meier (KM) plots of the cumulative incidence of double-blind IMP discontinuations due to any reason and due to AEs will be provided for the double-blind treatment period separately (see Section 2.5.4). A listing of these patients, along with the reason for discontinuation of treatment, study completion status and the reason for discontinuation study, will be provided.

For ABPM sub-study, the number of patients in each of the following categories will be summarized:

- Patients who consented to ABPM substudy.
- Patients not entering ABPM substudy and the reason for not entering.
- Patients who randomized and entered ABPM substudy (ie, ABPM substudy population, see Section 2.3.1.2).

Date of Issue: 15-Nov-2019 Lexicon Pharmaceuticals Protocol No. EFC14867 Covance Study ID: 000000155204

- Patients who completed ABPM substudy.
- Patients who discontinued ABPM substudy and the reason for discontinuation:
  - Adverse Event,
  - Study Terminated by Sponsor,
  - At patient's own request,
  - Lost to follow-up,
  - Poor compliance to Protocol,
  - Other.

For patients not entering ABPM substudy, percentages will be calculated using the number of patients consented to substudy as the denominator. All other categories of patients will be presented by treatment group and the percentages will be calculated using the number of patients randomized and entered substudy within each treatment group as the denominator. Reasons for ABPM substudy discontinuation will be supplied in tables giving numbers and percentages by treatment group. Patients prematurely discontinued the substudy, along with reasons for discontinuation, will also be listed. Patients who consented but did not enter ABPM substudy, along with reasons for not entering, will also be presented.

All important deviations including randomization and drug-dispensing irregularities will be summarized in tables giving numbers and percentages of deviations by randomized treatment group.

Additionally, the analysis populations for safety, efficacy, ABPM substudy, and pharmacokinetics defined in Section 2.3 will be summarized in a table by number of patients in the randomized population.

- Efficacy population: ITT population, completers population.
- Efficacy population for substudy: ABPM substudy population.
- Safety population.
- PK population.

# 2.2.1 Randomization and drug dispensing irregularities

Randomization and drug-dispensing irregularities occur whenever:

1. A randomization is not in accordance with the protocol-defined randomization method, such as a) an ineligible patient is randomized, b) a patient is randomized based on an incorrect stratum, c) a patient is randomized twice, or d) in a dynamic randomization scheme the treatment assignment is, in fact, not random, due to a computer program error.

OR

2. A patient is dispensed an IMP kit not allocated by the protocol-defined randomization, such as a) a patient at any time in the study is dispensed a different treatment kit than as

randomized (which may or may not contain the correct-as-randomized IMP), or b) a nonrandomized patient is treated with IMP reserved for randomized patients.

Randomization and drug-dispensing irregularities will be monitored throughout the study and reviewed on an ongoing basis.

All randomization and drug-dispensing irregularities will be documented in the clinical study report. If the number of irregularities is large enough to make a tabular summary useful, the irregularities will be categorized and summarized among randomized patients (number and percentages). Nonrandomized, treated patients will be described separately. Listings with additional, relevant details will be provided in appendices.

Randomization and drug-dispensing irregularities to be prospectively identified include but are not limited to:

#### Randomization and drug allocation irregularities

Kit dispensation without IRT transaction

Erroneous kit dispensation

Kit not available

Randomization by error

Patient randomized twice

Stratification error

Patient switched to another site

# 2.3 ANALYSIS POPULATIONS

Patients treated without being randomized will not be considered randomized and will not be included in any efficacy population.

The randomized population includes any patient who has been allocated to a randomized treatment regardless of whether the treatment kit was used.

For any patient randomized more than once, only the data associated with the first randomization will be used in any analysis population. The safety experience associated with any later randomization will be assessed separately.

The safety experience of patients treated and not randomized will be reported separately, and these patients will not be in the safety population.

#### 2.3.1 Efficacy populations

Efficacy analyses will be based on the treatment group allocated by the IRT according to the randomization schedule at randomization visit (as randomized), irrespective of the treatment actually received.

#### 2.3.1.1 Intent-to-treat population

Efficacy analyses will be based on the ITT population, defined as all randomized patients, irrespective of compliance with the study protocol and procedures. Patients will be analyzed for efficacy according to the treatment group to which they are randomized.

# 2.3.1.2 ABPM substudy population

ABPM efficacy analysis will be based on ABPM substudy population which defined as all randomized patients having:

- 1. Signed the informed consent for ABPM substudy
- 2. Baseline ABPM measurement at Visit 3A with Good Quality (see Appendix A)

# 2.3.1.3 Completers population

The completers population is a subset of the ITT population who complete the 26-week double-blind treatment period and without starting rescue therapy. A sensitivity analysis for noninferiority comparison will be conducted on this population.

#### 2.3.2 Safety population

Safety analyses will be based on the safety population, defined as all randomized patients who receive at least one dose or part of a dose of double-blind IMP (regardless of the amount of treatment administered). Patients will be analyzed according to the treatment actually received.

#### In addition:

- Nonrandomized but treated patients will not be part of the safety population, however, their safety data will be presented separately.
- Randomized patients for whom it is unclear whether they took the IMP will be included in the safety population as randomized.
- When a patient is exposed to both active treatment group and placebo, the patient will be analyzed in the corresponding active treatment group.
- When a patient is exposed to both sotagliflozin and empagliflozin, the patient will be analyzed in the sotagliflozin group.
- Randomized patients will be excluded from the safety population only if there is documented evidence (ie, all study dates recorded as no medication taken) that patients have not taken the study treatment. If a patient is dispensed double-blind IMP and is lost to follow-up without any documented evidence, the patient will be considered exposed.

#### 2.3.3 PK population

For PK analyses, the PK population is defined as all safety patients who contribute with at least 1 valid plasma concentration of sotagliflozin or its 3-O-glucuronide metabolite. The PK data will be analyzed according to the treatment actually received (see Section 2.3.2).

#### 2.4 STATISTICAL METHODS

#### 2.4.1 Demographics and baseline characteristics

Continuous data will be summarized using the number of observations available, mean, SD, median, minimum, and maximum for each treatment group. Categorical and ordinal data will be summarized using the count and percentage of patients in each treatment group.

Parameters will be summarized based on the randomized population analyzed in the treatment group to which they were randomized. Analyses for the safety population will be included in the appendices if the size of the safety population is different (>10%) from the size of that in the primary analysis population (ie, randomized patients) for any treatment group.

Parameters described in Section 2.1.1 will be summarized by treatment group and overall (pooled across treatment groups) using descriptive statistics.

P-values on the treatment difference for the demographic and baseline characteristic data will not be calculated.

In general, no specific description of the safety parameters will be provided at baseline. If relevant, the baseline values will be described along with each safety analysis.

In general, no specific description of the efficacy parameters will be provided at baseline. If relevant, the baseline values will be described along with each efficacy analysis.

#### 2.4.2 Prior or concomitant medications

The prior, concomitant and posttreatment medications will be presented in the randomized population for each treatment group (and overall for the summary of prior medications), using counts and percentages. No statistical test for the between-group difference will be performed.

Medications will be summarized by treatment group according to the WHO-DD dictionary, considering the first digit of the anatomical therapeutic chemical (ATC) class (anatomic category) and the first 3 digits of the ATC class (therapeutic category). A given medication may be classified in more than 1 ATC class. All ATC codes corresponding to a medication will be summarized, and a patient will be counted once in each ATC category (anatomic or therapeutic) linked to the medication. Therefore, a patient may be counted several times for the same medication.

Prior medications will be presented by anatomic and therapeutic categories and sorted by decreasing frequency of ATC based on the overall incidence across treatment groups. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

Concomitant and posttreatment medications will be presented by anatomic and therapeutic categories and sorted by decreasing frequency of ATC based on the incidence in the sotagliflozin 400mg group. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

# 2.4.3 Extent of investigational medicinal product exposure and compliance

The extent of IMP exposure and compliance will be assessed and summarized by actual treatment within the safety population (Section 2.3.2).

# 2.4.3.1 Extent of investigational medicinal product exposure

The extent of IMP exposure will be assessed by the duration of IMP exposure.

Duration of IMP exposure is defined as last dose date of double-blind IMP – first dose date of double-blind IMP + 1 day, regardless of unplanned intermittent discontinuations (see Section 2.5.3 for calculation in case of missing or incomplete data).

Duration of IMP exposure will be summarized descriptively as a quantitative variable (number of patients exposed, mean, SD, median, minimum, and maximum). In addition, duration of treatment exposure will also be summarized categorically by numbers and percentages for each of the following categories and cumulatively according to these categories:

- 1 to 28 days.
- 29 to 56 days.
- 57 to 84 days.
- 85 to 126 days.
- 127 to 182 days.
- >182 days.

Additionally, the cumulative duration of treatment exposure will be provided, defined as the sum of the duration of treatment exposure for all patients, and will be expressed in patient years.

Number and percentage of patients by final dose at the end of the treatment will also be presented by each treatment group.

# 2.4.3.2 Compliance

A given administration will be considered noncompliant if the patient did not take the planned dose of treatment as required by the protocol. No imputation will be made for patients with missing or incomplete data. Treatment compliance will be calculated and presented for sotagliflozin or matching placebo (Tablet) and empagliflozin or matching placebo (Capsule) separately by treatment group.

Percentage of compliance for a patient will be defined as the number of days that the patient was compliant to Capsule or Tablet, respectively, divided by the total number of days that the patient was planned to take IMP during the treatment epoch defined in Section 2.1.4 (ie, from the first date to the last date of double-blind IMP administration).

Above-planned dosing percentage for a patient will be defined as the number of days that the patient took a higher dose to Capsule or Tablet than planned, respectively, divided by the total number of days that the patient was planned to take during the treatment epoch.

Under-planned dosing percentage for a patient will be defined as the number of days that the patient took a lower dose to Capsule or Tablet than planned, respectively, divided by the total number of days that the patient was planned to take during the treatment epoch.
Treatment compliance, above-planned, and under-planned dosing percentages will be summarized for Capsule and Tablet separately and descriptively as quantitative variables (number, mean, SD, median, minimum, and maximum). The percentage of patients whose compliance is <80% will be summarized. In addition, numbers and percentages of patients with at least 1 day above-planned dose will be provided, as well as numbers and percentages of patients with (0, 20%], and >20% of days under-planned dose.

Cases of overdose (see study protocol for further details) will constitute AEs/SAEs and be analyzed as such. More generally, dosing irregularities will be listed in Section 2.2.1.

# 2.4.4 Analyses of efficacy endpoints

Efficacy analyses will be performed on the ITT population using the efficacy assessments collected during the study, including those obtained after IMP discontinuation or introduction of rescue therapy, unless otherwise specified.

Missing data for efficacy analyses is identified through steps described in Section 2.5.4.

# 2.4.4.1 Analysis of primary efficacy endpoint

The statistical test will be two-sided tests at a nominal 5% significance level.

# Primary analysis

The primary efficacy endpoint of change in HbA1c from baseline to Week 26 will be analyzed by an Analysis of Covariance (ANCOVA) model using HbA1c values measured at baseline and Week 26 (observed or imputed). The missing data at endpoint will be imputed by multiple imputation (MI) methods as detailed below. To be concise, the following texts related to imputation are generalized to accommodate primary as well as continuous secondary efficacy endpoints.

Missing endpoint data at Week 26 (or Week 12 for SBP) visit will be imputed using a model built separately in each treatment group and estimated from the patients in the same treatment group who prematurely discontinue the IMP before the Week 26 (or Week 12 for SBP) visit but have the measurement for the endpoint (ie, retrieved dropouts). The imputation model will include the randomization strata and the corresponding baseline value. In cases of non-convergence during the imputations, the offending stratum will be identified and then will be dropped from the model. Considering that the number of retrieved dropout patients in each treatment group is expected to be small, a simple imputation model based on regression will be used with baseline measurement included as the predictor. This will serve as the primary model of imputation for missing data should sampling criteria be satisfied (see below).

An alternative (back-up) imputation method will be used if the number of patients who prematurely discontinue the IMP before the Week 26 (or Week 12 for SBP) visit but have the measurement for the endpoint is < 5 in any treatment groups (ie, insufficient number of retrieved

dropouts to support the imputation method described above). This criterion will be assessed for each primary or continuous secondary efficacy endpoint.

In the back-up imputation method, missing post-baseline endpoint values at Week 26 (or Week 12 for SBP) will be imputed by the washout Multiple Imputation (MI) method under the missing not at random (MNAR) framework.

Missing endpoint data at the Week 26 (or Week 12 for SBP) in all treatment groups (sotagliflozin 400 mg, empagliflozin 25 mg and placebo) are imputed from a model estimated from patients in the placebo group who have the endpoint data available.

For patients in the sotagliflozin 400 mg and empagliflozin 25 mg groups with missing data at Week 26 (or Week 12 for SBP), their missing values will be imputed using observed baseline and the observed primary endpoint data from placebo completers; no intermittent values from either placebo or the active treatment groups will be used.

For placebo patients, missing data will be imputed based on the placebo group data. Intermittent observed values will be used while imputing missing values at Week 26 (or Week 12 for SBP). In cases that a non-monotone missing data pattern occurs at the intermediate visits, these data points will be first imputed in the placebo group using the Markov Chain Monte Carlo (MCMC) option in PROC MI to achieve a monotone missing pattern for all placebo patients. The Week 26 (or Week 12 for SBP) endpoint values will be subsequently imputed from the multiple copies of the original dataset where each copy will have a monotone missing pattern.

The imputation models for the washout MI method will include the randomization strata and the corresponding baseline value. Missing data will be imputed using the regression method.

In cases of non-convergence during the imputations, especially for the MCMC application in the placebo non-monotone datasets, graphical measures (eg, trace and autocorrelation plots) will be used to identify the offending variable and once detected, that variable(s) will be dropped from the model and the imputations will be re-run. These re-run models will use the same seed number and number of imputations as used in the original models.

Using either imputation method, missing endpoint data will be imputed 2000 times to generate multiple data sets with complete data. Other details of the imputation procedures such as the seed number and sort ordering are specified in the SAS programs. The HbA1c change from baseline to Week 26 (or Week 12 for SBP) will be derived from observed and imputed HbA1c values at Week 26 (or Week 12 for SBP). Each of the completed datasets after the imputation will be analyzed using the Analysis of Covariance (ANCOVA) model with treatment groups (sotagliflozin 400 mg, empagliflozin 25 mg and placebo), randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at screening (Yes, No), randomization stratum of SBP (<130 mmHg, ≥130 mmHg), and country as fixed factors, and baseline HbA1c value as a covariate. Results from each analysis will be combined using Rubin's formula, to provide the adjusted mean change in HbA1c from Baseline to Week 26 (or Week 12 for SBP) for each treatment group, as well as the between-group difference (comparing sotagliflozin 400 mg versus placebo) and its associated 95% confidence interval (CI).

# Sensitivity analyses

Tipping point analysis based on the same MI method as applied to the primary analysis will be performed to examine the robustness of the results from the primary analysis. Patients who were randomized to sotagliflozin 400 mg group and had no HbA1c data at Week 26 will be given a penalty. The penalty will be gradually increased to evaluate at which level the conclusion of the analyses in terms of statistical significance is changed. The tipping point is the penalty level, at which the magnitude of efficacy reduction in patients without HbA1c data at Week 26 creates a shift in the treatment effect of sotagliflozin 400 mg from being statistically significantly better than placebo to a non-statistically significant effect. LS mean difference between sotagliflozin 400 mg and placebo and its associated p-value for superiority will be provided for each penalty level. The steps to perform the tipping point analysis are as follows:

- 1. Missing data will be imputed using the same MI method as applied to the primary analysis,
- 2. The imputed HbA1c value at Week 26 in the sotagliflozin 400 mg group will be penalized by adding a penalty  $\delta$  (eg,  $\delta$  = 0.1%) in each complete dataset,
- 3. Change from baseline at Week 26 in HbA1c will be analyzed using the same ANCOVA model as specified in the primary analysis in each complete dataset,
- 4. Results will be combined across complete datasets using Rubin's formula,
- 5. For superiority of sotagliflozin 400 mg versus placebo on HbA1c reduction, steps 2 to 4 will be repeated with incremental penalty at  $\delta$  (ie,  $\delta$ ,  $\delta$ ,  $\delta$ ,  $\delta$ ,  $\delta$ , .....) until the p-value for treatment effect of sotagliflozin 400 mg compared to placebo estimated in Step 4 is >0.05.
- 6. For noninferiority of sotagliflozin 400 mg versus empagliflozin 25 mg on HbA1c reduction, Steps 2 to 4 will be repeated with incremental penalty at δ (ie, δ, 2δ, 3δ, .....) until the upper bound of the 2-sided 95% CI for the adjusted mean difference is >0.3. The range of penalty values will include the non-inferiority margin of 0.3% to evaluate bias toward the null.

The tipping point analysis will be performed on the ITT population and completer's population. The tipping point analysis will be performed for the primary variable only if that variable (change from baseline to Week 26 in HbA1c comparing sotagliflozin 400 mg versus placebo) is statistically significant at  $\alpha = 0.05$  (2-sided). Similarly, the tipping point analysis will be conducted for the sotaglifozin 400 mg versus empaglifozin 25 mg non-inferiority endpoint only if the primary efficacy endpoint analysis yields a statistically significant finding and the upper bound of the 2-sided 95% CI associated with the non-inferiority test is < 0.3%.

In addition to the tipping point analyses, if the retrieved dropout imputation is applied to the primary analysis, the analysis based on the washout imputation method (ie, the backup imputation method) will be presented as a sensitivity analysis.

Patients in this study have undergone sampling for plasma levels of sotagliflozin and its main active metabolite in order to perform population PK analysis. Patients may be identified who have no detectable levels of active study drug or metabolite in their samples (ie, Below Lower Limit of

Quantification or BLLOQ). When sample analysis has been completed and the study has been unblinded, explanations for some of these patients may be found: known non-compliance or sampling occurring after treatment had been discontinued. In other cases, drug intake history relative to the randomization assignment may not be fully explained. The ITT-based analyses specified in this document provides for a conservative assessment of the efficacy data should patients have been subjected to these unexplained non-compliance findings or PK 'anomalies'. To provide a broader perspective on the impact of these apparent errors in compliance, additional sensitivity analyses of the primary efficacy endpoint and continuous efficacy endpoints may be conducted. The need to perform such analyses, their specifics, and results will be provided in the Clinical Study Report (CSR), if applicable. The analysis methods applied to the patient subpopulations defined by the occurrence of the PK anomalies (eg., exclusion of patients with PK anomalies from the ITT dataset) will include the ANCOVA model using the retrieved dropout and/or washout MI methods previously specified in this section.

# Assessment of treatment effect by subgroup

Descriptive analyses will be performed on the primary endpoint to summarize the treatment effects across subgroups defined by the following baseline or screening factors:

- Race (White, Black or African American, Asian, Other) (any race groups with fewer than 5 patients may be combined with "Other" category as appropriate).
- Ethnicity (Hispanic, Not Hispanic).
- Age group ( $<50, \ge 50$  to  $<65, \ge 65$  years) (any category with fewer than 5 patients may be combined with another category as appropriate).
- Gender (Male, Female).
- Baseline BMI level ( $<30, \ge 30 \text{ kg/m}^2$ ).
- Baseline HbA1c ( $\leq 8.5\%$ , > 8.5%).
- Metformin use at Screening (Yes, No).
- Baseline mean SBP (<130 mmHg, ≥130 mmHg).
- Baseline eGFR (≥30 to <60 mL/min/1.73m<sup>2</sup> [Moderate decrease in GFR], ≥60 to <90 mL/min/1.73m<sup>2</sup> [Mild decrease in GFR], and ≥90 mL/min/1.73m<sup>2</sup> [Normal]).
- Duration of diabetes ( $<10, \ge 10$  years).
- Country.

The treatment effects (sotagliflozin 400 mg versus placebo) across the subgroups defined for each of these factors will be estimated for the change from Baseline to Week 26 in HbA1c in the ITT population, and using the retrieved dropout method if there are at least 5 patients in each study treatment group who discontinued but have the endpoint. Otherwise, the washout imputation method will be used. The ANCOVA model will include treatment groups

(sotagliflozin 400 mg, empagliflozin 25 mg, placebo), randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at screening (Yes, No), randomization stratum of SBP at screening (<130 mmHg, ≥130 mmHg), subgroup factor, treatment-by-subgroup factor, and country as fixed factors and using baseline HbA1c value as a covariate. The adjusted estimates of treatment mean differences (sotagliflozin 400 mg versus placebo) with SE and 95% CIs will be provided as appropriate across the subgroups. A graphical presentation of the results (ie, forest plot) will also be provided.

In the case that the subgroup factor is identical or similar to a randomization strata factor (eg, baseline HbA1c, metformin use at screening, or baseline mean SBP category), only the subgroup factor (as a single factor or an interaction term) will be included in the model in order to avoid the issue of collinearity in the analysis. The corresponding strata factor will not be included in the model.

# Summary statistics at scheduled visits

Summary statistics (for screening value, baseline value, observed post-baseline value and its changes from baseline) at scheduled visits will be provided for each treatment group. The summary will include the number of observations, mean, SD, SE, minimum, median, and maximum. Graphical presentations will also be used to examine trends over time using mean values (±SE) and mean changes from baseline (±SE) at each of the scheduled visits.

Similar presentations will be provided excluding measurements after rescue therapy during the 26-week double-blind treatment period.

# 2.4.4.2 Analyses of secondary efficacy endpoints

For continuous secondary efficacy parameters (Section 2.1.3) with missing data at baseline, missing baseline data will be imputed using MI under the missing at random (MAR) assumption. Missing data at baseline will be imputed using regression method that includes randomization stratum of HbA1c ( $\leq$ 8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), randomization stratum of SBP (<130 mmHg,  $\geq$ 130 mmHg), and baseline value in the imputation model .

Each continuous secondary efficacy endpoint (Section 2.1.3) will be analyzed using a similar ANCOVA model including the measurements at baseline and endpoint (observed or imputed). The missing data at endpoint will be imputed by the retrieved dropouts if there are at least 5 patients in each study treatment group who discontinued but have the endpoint. Otherwise, the washout imputation method will be used. After the imputation, each of the complete datasets will be analyzed by an ANCOVA model.

The ANCOVA model will include treatment groups (sotagliflozin 400 mg, empagliflozin 25 mg and placebo), randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), randomization stratum of SBP (<130 mmHg, ≥130 mmHg), and country as fixed effects, and the corresponding baseline secondary endpoint

value as a covariate. For the analysis of SBP in patients with baseline SBP ≥130 mmHg, the randomization stratum of SBP will not be included. Results from each complete dataset will be combined using Rubin's formula to provide the adjusted mean change from Baseline to Week 26 (or Week 12 for SBP) for each treatment group, as well as the between-group differences and the 95% CIs for the differences.

For all continuous secondary endpoints, summary statistics at scheduled visits will be provided for each treatment group. The summary will include the number of observations, mean, SD, SE, minimum, median, and maximum. Graphical presentations will also be used to examine trends over time using mean values ( $\pm$ SE) and mean changes from baseline ( $\pm$ SE) at each of the scheduled visits. In addition, SBP will be summarized descriptively at each visit for those patients with baseline SBP  $\geq$ 140 mmHg.

The categorical secondary efficacy variables of HbA1c <6.5%, <7% at Week 26 will be analyzed respectively using a Cochran-Mantel-Haenszel (CMH) method stratified by randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), and randomization stratum of SBP (<130 mmHg, ≥130 mmHg). The proportion in each treatment group will be provided, as well as the difference of proportions between sotagliflozin 400 mg and placebo with associated 2-sided 95% CI. For HbA1c responders at Week 26 (<6.5%, <7% respectively), all values at Week 26 will be used to determine whether a patient is a responder or not, even if they are measured after IMP discontinuation or rescue medication use. Patients who have no HbA1c measurement at Week 26 will be treated as non-responders. Summary tables and graphs will also be provided by treatment group at scheduled visits.

For between-group comparison, a sensitivity analysis will be performed respectively for HbA1c <6.5% responder analysis by excluding patients whose HbA1c values at baseline are <6.5%, and for HbA1c <7% responder analysis by excluding patients whose HbA1c values at baseline are <7% using the same CMH test mentioned above. Similarly, by-visit summary may also be provided excluding those patients.

#### Noninferiority on HbA1c reduction

Tipping point analysis, described in Section 2.4.4.1, will be performed to examine the robustness of the noninferiority of sotagliflozin 400 mg versus empagliflozin 25 mg on HbA1c reduction using the same imputation method and ANCOVA model as described in Section 2.4.4.1. LS mean difference between sotagliflozin 400 mg and empagliflozin 25 mg will be provided for each penalty level. The tipping point analysis will be performed only if the primary endpoint analysis is positive with an observed p-value  $\leq 0.05$  and the secondary endpoint analysis of the noninferiority of sotagliflozin 400 mg versus empagliflozin 25 mg on HbA1c reduction at Week 26 is positive; ie, the upper bound of the 2-sided 95% CI is  $\leq 0.3\%$ .

The treatment effects (sotagliflozin 400 mg versus empagliflozin 25 mg) across the subgroups (defined in Section 2.4.4.1) will be estimated for the change from Baseline to Week 26 in HbA1c in the ITT population, and using the same approach described in Section 2.4.4.1. The adjusted estimates of treatment mean differences (sotagliflozin 400 mg versus empagliflozin 25 mg) with

SE and 95% CIs will be provided as appropriate across the subgroups. A graphical presentation of the results (ie, forest plot) will also be provided.

A sensitivity analysis will be conducted with the treatment completers (ie, all patients who complete the 26-week double-blind treatment period and do not start rescue therapy) for noninferiority of sotagliflozin 400 mg versus empagliflozin 25 mg on HbA1c reduction using the same ANCOVA model described in Section 2.4.4.1. The washout imputation method will be used, where missing endpoint data in all treatment groups are imputed from a model estimated from patients in the placebo group who have the endpoint data available. The imputation model will include the randomization strata and the corresponding baseline value. Missing data will be imputed using the regression method.

## 2.4.4.3 Analyses of other efficacy endpoints

The analysis of other endpoints (see Section 2.1.3) will be descriptive with no formal testing. Summary statistics at scheduled visits based on observed value will be provided by each treatment group. Graphical presentations will also be used to illustrate trends over time as appropriate. The exception to this plan is for UGE, urine GCR, and the originally listed secondary endpoints recategorized as 'Other' endpoints (see Section 2.4.4.5). The sotagliflozin 400 mg versus placebo and sotagliflozin 400 mg versus empagliflozin 25 mg comparisons for these variables will be subjected to statistical analyses as described in Section 2.4.4.2.

The number (%) of patients who used rescue therapy and a KM curve for the time to first rescue therapy will be provided by treatment group. A list of patients who used rescue therapy will also be provided (see Section 2.5.4).

Urine ACR will be log-transformed at patient level. Summary statistics of urine ACR in log scale will then be calculated for each treatment group at each visit and back-transformed to provide the geometric mean and its associated percent change of urine ACR from baseline.

Shift tables will be provided for urine ACR at Week 26 using the pre-defined categories. That is, the number (%) of patients with progression from one category at baseline to another category at Week 26 will be provided by treatment group. The pre-defined categories are, for urine ACR, <30 mg/g creatinine [Normal], ≥30 to <300 mg/g creatinine [Microalbuminuria], and ≥300 mg/g creatinine [Macroalbuminuria].

The analysis of the 2-hour PPG endpoint will be based on a Time 0 adjusted value (ie, the 2-hour PPG value minus the Time 0 value, FPG sample) at both the Baseline and Week 26 time points. These Time 0 adjusted values will be used to derive the Week 26 minus Baseline scores, which will serve as the measure of interest for comparative purposes.

# 2.4.4.4 Analysis of ABPM substudy efficacy endpoints

Analyses of ABPM substudy efficacy endpoints will be performed on the ABPM population using all assessment collected up to Week 26. All ABPM substudy efficacy endpoints will be

summarized by descriptive statistics at scheduled visits (Baseline (Visit 3A, Week -1), Visit 6A (Week 12), and Visit 8A (Week 26)). The descriptive statistics will include number, mean, standard deviation, Q1, Q3, minimum, maximum. In addition, analyses will be done for those patients with baseline Mean 24-hour SBP ≥130 mmHg and those patients with baseline Mean 24-hour SBP <130 mmHg separately.

Please refer to Appendix A and Appendix B for ABPM substudy efficacy variable derivation.

## 2.4.4.5 Multiplicity issues

To control for the family-wise type I error, a fixed-sequence procedure will be applied.

Once the primary hypothesis (superiority of the change from Baseline to Week 26 in HbA1c comparing sotagliflozin 400 mg versus placebo) is statistically significant for the primary efficacy endpoint, the following secondary hypothesis based on change from Baseline scores will be tested in the following prioritized order:

1. The noninferiority of sotagliflozin 400 mg versus empagliflozin 25 mg on HbA1c reduction at Week 26,

The superiority of sotagliflozin 400 mg versus placebo on:

- 2. 2-hour PPG reduction at Week 26,
- 3. Body weight reduction at Week 26,
- 4. Sitting SBP reduction at Week 12 in patients with Baseline SBP ≥130 mmHg,

The superiority of sotagliflozin 400 mg versus empagliflozin 25 mg on:

- 5. 2-hour PPG reduction at Week 26,
- 6. HbA1c reduction at Week 26,
- 7. Sitting SBP reduction at Week 12 in patients with Baseline SBP ≥130 mmHg,
- 8. Sitting SBP reduction at Week 12.

If any hypothesis is found to be not statistically significant, the testing procedure will be stopped and the following hypotheses will not be tested. The noninferiority hypothesis will be declared significant if the upper bound of the 2-sided 95% CI for the adjusted mean difference is <0.3. The superiority hypothesis will be declared statistically significant at  $\alpha = 0.05$  (2-sided). This hierarchy differs from the ordering provided in the study protocol and that is likewise reflected in Section 1.2.2 of this SAP. The Sponsor elected to modify the contents/testing order to maximize

the number of rejected null hypotheses. These modifications were made before unblinding of the database.

The secondary endpoints omitted from the original testing hierarchy will still be subjected to the analysis methods specified in Section 2.4.4.2. However, these variables will be labeled as 'Other' endpoints and not secondary endpoints.

No multiplicity adjustment will be made on efficacy variables other than those mentioned above.

# 2.4.5 Analyses of safety data

The summary of safety results will be presented by treatment group.

The "observation period" defined in Section 2.1.4 is applicable in all safety analyses for the classification of AEs, determination of treatment-emergent Potentially Clinically Significant Abnormality (PCSA) values and the last on-treatment value for the laboratory, vital sign and ECG.

#### General common rules

All safety analyses will be performed on the safety population as defined in Section 2.3.2, unless otherwise specified, using the following common rules:

- Safety data in patients who do not belong to the safety population (eg, exposed but not randomized) will be listed separately.
- The baseline value (with the exception of serum creatinine and eGFR) is defined as the last available value before the first dose of double-blind IMP. For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP.
- PCSA values are defined as abnormal values considered medically important by the Sponsor according to predefined criteria/thresholds based on literature review and defined by the Sponsor for clinical laboratory tests, vital signs, and ECG Appendix C.
- PCSA criteria will determine which patients had at least 1 PCSA during the TEAE period, taking into account all evaluations performed during the TEAE period, including nonscheduled or repeated evaluations. The number of all such patients will be the numerator for the treatment-emergent PCSA percentage.
- The treatment-emergent PCSA denominator by group for a given parameter will be based on the number of patients assessed for that given parameter during the TEAE period by treatment group in the safety population.
- For laboratory parameters cited in the protocol as efficacy endpoints (including HbA1c and plasma glucose etc.), PCSA summaries will not be provided. These parameters will be summarized in efficacy Section 2.4.4. For creatinine and eGFR, PCSA summaries will be presented in safety Section 2.4.5 while descriptive summaries in efficacy Section 2.4.4.

• For quantitative safety parameters based on central laboratory/reading measurements, descriptive statistics will be used to summarize results and change from baseline values by visit and treatment group. Summaries will include the last on-treatment value. The last ontreatment value is commonly defined as the value collected at the same day/time of the last administration of IMP. If this value is missing, this last on-treatment value will be the closest value prior to the last dose administration.

- The analysis of the safety variables will be essentially descriptive and no systematic testing is planned. Relative risks versus placebo and empagliflozin, and their 95% CIs may be provided, if relevant.
- Selected safety analyses will be summarized by age, gender, racial subgroups, and other pertinent subgroups (see details in Section 2.4.5.1 and Section 2.4.5.2).

# 2.4.5.1 Analyses of hypoglycemia

Analyses of hypoglycemia will be performed on the TEAE period as defined in Section 2.1.4. Hypoglycemia will be classified as severe hypoglycemia, documented symptomatic hypoglycemia, asymptomatic hypoglycemia, probable symptomatic hypoglycemia or relative hypoglycemia (see Section 2.1.4.1).

The number (%) of patients with any hypoglycemia, severe hypoglycemia and documented symptomatic hypoglycemia will be summarized respectively by treatment group during the TEAE period, as well as the incidence rate in patient years. Two types of incidence rates will be presented: the number of patients with at least 1 event per 100 patient-years (calculated as the number of patients with at least 1 event / total exposure in 100 patient-years), and the number of events per 100 patient-years (calculated as the total number of events / total exposure in 100 patient-years). Note: here exposure (in days) is the duration of TEAE period, ie, duration of IMP treatment in days +1 (see Section 2.1.4).

The summary of frequency and incidence rate in patient years for severe hypoglycemia or documented symptomatic hypoglycemia will be provided as appropriate by gender (Male, Female), age group ( $<50, \ge 50$  to  $<65, \ge 65$  years), race (White, Black or African American, Asian, Other) and metformin use at Screening (Yes, No).

A KM curve will also be provided by treatment group for the time to first severe hypoglycemia or documented symptomatic hypoglycemia during the TEAE period (see Section 2.5.4).

Documented symptomatic hypoglycemia maybe presented by  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL) and ( $\leq$ 3.0 mmol/L ( $\leq$ 54 mg/dL) respectively, as appropriate.

A listing of patients for all events reported on the dedicated e-CRF "Hypoglycemic event information" page will be provided with each category flagged (ie, severe hypoglycemia,

documented symptomatic hypoglycemia, asymptomatic hypoglycemia, probable symptomatic hypoglycemia and relative hypoglycemia).

## 2.4.5.2 Analyses of adverse events

#### **Generalities**

The primary focus of adverse event reporting will be on treatment-emergent adverse events. Pretreatment and posttreatment adverse events will be described separately.

If an adverse event date/time of onset (occurrence, worsening, or becoming serious) is incomplete, an imputation algorithm will be used to classify the adverse event as pretreatment, treatment-emergent, or posttreatment. The algorithm for imputing date/time of onset will be conservative and will classify an adverse event as treatment emergent unless there is definitive information to determine it is pretreatment or posttreatment. Details on classification of adverse events with missing or partial onset dates are provided in Section 2.5.3.

Adverse event incidence tables will be presented by SOC, HLGT, HLT, and PT, sorted by the internationally agreed order for SOCs and alphabetic order for HLGT, HLT and PT within a SOC, the number (n) and percentage (%) of patients experiencing an adverse event. Multiple occurrences of the same event in the same patient will be counted only once in the tables within a treatment phase. The denominator for computation of percentages is the safety population within each treatment group.

Sorting within tables ensures the same presentation for the set of all adverse events within the observation period (pretreatment, treatment-emergent, and posttreatment). For that purpose, the table of all treatment-emergent adverse events presented by primary SOC and PT (sorted by the internationally agreed SOC order and decreasing frequency of PTs within SOCs in the sotagliflozin 400 mg group) will define the presentation order for all other similar tables unless otherwise specified. In case of equal frequency regarding PTs, alphabetical order will be used.

#### Analysis of all treatment-emergent adverse events

The following treatment-emergent adverse event summaries will be generated for the safety population.

- Overview of treatment-emergent adverse events, summarizing number (%) of patients with any:
  - TEAE,
  - Serious TEAE,
  - TEAE leading to death,
  - TEAE leading to permanent treatment discontinuation.
- All treatment-emergent adverse events by primary SOC, showing number (%) of patients
  with at least 1 treatment-emergent adverse event, sorted by internationally agreed order of
  primary system organ class.

• All treatment-emergent adverse event by primary SOC, HLGT, HLT, and PT, showing number (%) of patients with at least 1 treatment-emergent adverse event sorted by the SOC internationally agreed order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.

- Number (%) of patients experiencing TEAE(s) presented by PT, sorted by decreasing incidence of PT in the sotagliflozin 400 mg group.
- All treatment-emergent adverse events by primary SOC and PT, showing the number (%) of patients with at least 1 treatment-emergent adverse event, sorted by the internationally agreed SOC order and by decreasing incidence of PTs within each SOC in the sotagliflozin 400 mg group. This sorting order will be applied to all other similar tables, unless otherwise specified.
- All treatment-emergent adverse events regardless of relationship and related to IMP by primary SOC, HLGT, HLT and PT, showing the number (%) of patients with at least 1 treatment-emergent adverse event, sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.
- All treatment-emergent adverse events by maximal severity, presented by primary SOC and PT, showing the number (%) of patients with at least 1 treatment-emergent adverse event by severity (ie, mild, moderate, or severe), sorted by the sorting order defined above.
- Common TEAEs (PTs with an incidence ≥2% in any treatment group) by primary SOC, HLGT, HLT, and PT, sorted by internationally agreed order of SOCs. The other levels (HLGT, HLT, PT) will be presented in alphabetic order.
- Common TEAEs (PTs with an incidence ≥2% in any treatment group) will be provided as appropriate by primary SOC and PT and by demographic factors including gender (Male, Female), age group (<50, ≥50 to <65, ≥65 years of age), race (White, Black or African American, Asian, other), baseline SBP category (<130 mmHg, ≥130 mmHg), and baseline eGFR category (≥30 to <60 mL/min/1.73m² [Moderate decrease in GFR], ≥60 to <90 mL/min/1.73m² [Mild decrease in GFR], and ≥90 mL/min/1.73m² [Normal]). SOC will be sorted by internationally agreed order and the PT by decreasing incidence within each SOC in the sotagliflozin 400 mg group, as described above.
- TEAEs (PTs with an incidence ≥5% in any treatment group) by primary SOC, HLGT, HLT, and PT, sorted by internationally agreed order of SOCs. The other levels (HLGT, HLT, PT) will be presented in alphabetic order.

# Analysis of all treatment emergent serious adverse event(s)

- All treatment-emergent SAE by primary SOC, HLGT, HLT, and PT, showing the number (%) of patients with at least 1 serious treatment-emergent adverse event, sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.
- All treatment-emergent SAE regardless of relationship and related to IMP, by primary SOC, HLGT, HLT, and PT, showing the number (%) of patients with at least 1 serious

treatment-emergent adverse event, sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.

## Analysis of all treatment-emergent adverse event(s) leading to treatment discontinuation

• All treatment-emergent adverse events leading to treatment discontinuation, by primary SOC, HLGT, HLT, and PT, showing the number (%) of patients sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.

# Analysis of adverse events of special interest

Pregnancy and overdose will be included in overall AE summaries if any are reported. ALT increase >3 x ULN is included in laboratory PCSA summary if any.

In addition, the number (%) of patients with an AESI will be summarized by PT and by treatment group. Corresponding listings will be provided as appropriately.

# Analysis of events of special interest

# CV events, bone fracture and DKA

For EOSIs that are adjudicated (ie, deaths, myocardial infarction, stroke, and unstable angina requiring hospitalization, heart failure requiring hospitalization, bone fracture, and diabetic ketoacidosis), the number (%) of patients with an EOSI positively adjudicated by CEC will be summarized by treatment group. All EOSIs sent for adjudication and/or reported by the investigators in the specific AE forms will be listed along with the adjudication outcome.

#### Renal events

For the EOSI renal events where selected events are adjudicated, the number (%) of patients with any renal events identified in Table 3 in Section 2.1.4.2 will be summarized by treatment group.

The following renal events will be listed along with the adjudication outcome if applicable, including events,

- i. recorded in e-CRF "GFR decrease",
- ii. recorded in e-CRF "Renal Event Dialysis",
- iii. identified as "Renal transplant" in e-CRF "Other procedure".

Renal death will be part of all deaths specified above.

#### Other EOSIs

For EOSIs that are not adjudicated, the number (%) of patients with at least one event will be summarized by treatment group and by PT (as identified in Table 3 Section 2.1.4.2).

Severe hypoglycemia will be included in the summary of hypoglycemia (See Section 2.4.5.1).

AE leading to an amputation is described in the section below.

# Analysis of Amputation

The number (%) of patients with amputation will be summarized by treatment group and by PT and LLT during the study (ie, regardless of on- or post-treatment). Amputation is a procedure recorded in e-CRF form "Other Procedures related to Amputation". Patients who had a procedure related to amputation will be listed.

The number (%) of patients with an "AE leading to an amputation" will be summarized by treatment group and by PT. The "AE leading to an amputation" is determined by the AE identifier recorded in e-CRF "Other Procedures related to Amputation" when "AE correction" is chosen as the reason for the amputation procedure.

In addition, the number (%) of patients with an "AE potentially leading to an amputation" will be summarized by treatment group and by PT (as identified in Table 3 in Section 2.1.4.2; these PTs in Table 3 were requested by the European Medicines Agency/ Pharmacovigilance Risk Assessment Committee[EMA/PRAC] Assessment Report 9 February 2017). Associated list will be provided as well, with patients who had an amputation procedure flagged. "AE potentially leading to an amputation" represents the condition that may potentially lead to the amputation procedure, but not in all cases an amputation has occurred (as per the EMA/PRAC request).

## Analysis of pretreatment and posttreatment adverse events

- All pretreatment adverse events by primary SOC and PT, showing the number (%) of
  patients with at least 1 pretreatment adverse event, sorted by the internationally agreed
  SOC order and decreasing incidence of PTs within each SOC in the sotagliflozin
  400 mg group.
- All posttreatment adverse events by primary SOC and PT, showing the number (%) of patients with at least 1 posttreatment adverse event, sorted by the internationally agreed SOC order and decreasing incidence of PTs within each SOC in the sotagliflozin 400 mg group.

# Listings

Supportive AE listings will be provided for all AEs, SAEs, death, AEs leading to treatment discontinuation and/or death, and EOSI as appropriate. Listing of all AEs, SAEs and AEs leading to treatment discontinuation and/or death will include at least the following information, sorted by treatment, patient identification, and onset date: treatment, patient identification, country, age, gender, race, BMI, primary SOC, PT, reported term, onset date, study day (relative day to the start date of double-blind treatment), AE duration, duration of exposure, intensity, corrective treatment, action taken with IMP, date of treatment discontinuation (if relevant), relationship to IMP (sotagliflozin/matching placebo tablet and empagliflozin/matching capsule) or NIMP, outcome, date of death (if any), seriousness, seriousness criteria, and AE status ("E" for a TEAE; and "P" for an on-study post-treatment AE).

## 2.4.5.3 Deaths

The following summaries of deaths will be generated.

- Number (%) of patients who died by study period (on-study, on-treatment, post-study).
- Deaths in nonrandomized patients or randomized but not treated patients.
- Treatment-emergent adverse events leading to death (death as an outcome on the adverse event e-CRF page as reported by the Investigator) by primary SOC, HLGT, HLT, and PT showing number (%) of patients sorted by internationally agreed SOC order, with HLGT, HLT, and PT presented in alphabetical order within each SOC.

# 2.4.5.4 Analyses of laboratory variables

Laboratory parameters will be grouped and summarized by biological function as described in Section 2.1.4.4.

The summary statistics (including number, mean, median, Q1, Q3, standard deviation, minimum and maximum) of all laboratory variables (central laboratory values and changes from baseline) will be calculated for each applicable visit or study assessment (screening, baseline, postbaseline time point, last on-treatment value) by treatment group.

The incidence of PCSAs (list provided in Appendix D) at any time during the TEAE period will be summarized for each laboratory test by biological function and treatment group whatever the baseline level and/or according to the following baseline status categories:

- Normal/missing.
- Abnormal according to PCSA criterion or criteria.

For parameters for which no PCSA criteria are defined, similar table(s) using the normal range will be provided.

All measurements collected during the TEAE period, including values from unscheduled visits, will be considered for the PCSA summaries. These summaries will include patients in the safety population who have at least 1 assessment performed during the TEAE period. When a PCSA definition involves a change from baseline value, patients must also have a baseline value to be included in the summaries, and when required by the definition of the abnormality, patients must also have available laboratory normal ranges.

A listing of patients with at least 1 post-baseline PCSA (or out of normal range when no PCSA criterion is defined) will be provided and will display the entire patients' profile across time for all parameters belonging to the corresponding biological function. Individual data listings will include the following flags when applicable:

- Baseline values will be flagged "B".
- Normal laboratory ranges, available for most laboratory parameters, will be identified as ULN and LLN. Baseline, last on-treatment value, and individual data will be flagged "L" if the value is below the LLN and will be flagged "H" if it is above the ULN.

• Laboratory PCSA criteria will be used for the corresponding laboratory parameters. Values reaching a PCSA limit will be flagged (+, ++, -, or -- depending upon the direction and level of the abnormality). Flags for WBC and differential counts will be determined using data expressed in international units.

For parameters whose PCSA criteria are multiples of the ULN, the parameter's value will also be expressed as a multiple of the ULN in the individual data provided.

# Drug-induced liver injury

The liver function tests, namely AST, ALT, alkaline phosphatase, and total bilirubin, are used to assess possible drug-induced liver toxicity. The proportion of patients with PCSA values at any postbaseline visit by baseline status will be displayed by treatment group for each parameter. The proportion of patients with PCSA values at any postbaseline visit will also be displayed by duration of exposure for each treatment group (only if a tabulation summary is necessary).

Listing of possible Hy's law cases identified by treatment group (eg, patients with any elevated ALT>3 x ULN, and associated with an increase in bilirubin ≥2 x ULN) with ALT, AST, alkaline phosphatase, total bilirubin, and the following complementary parameters (if available): conjugated bilirubin and prothrombin time/international normalized ratio, creatine phosphokinase, serum creatinine, complete blood count, anti-HAV IgM, anti-HBc IgM, anti-HCV and HCV RNA, anti-CMV IgM and anti-HEV IgM antibodies, auto-antibodies: anti-nuclear, anti-DNA, anti-smooth muscle, Epstein-Barr virus, herpes viruses, and anti-LKM.

# 2.4.5.5 Analyses of vital sign variables

The summary statistics (including number, mean, median, Q1, Q3, standard deviation, minimum and maximum) of heart rate, temperature and respiratory rate (observed values or mean of observed values, and changes from baseline) will be calculated for each applicable visit or study assessment (baseline, post-baseline time points, last on-treatment value) by treatment group.

The incidence of PCSAs at any time during the TEAE period will be summarized by treatment group for SBP, DBP and HR. All measurements collected during the TEAE period, including values from unscheduled visits, will be considered for the PCSA summaries. The summaries will include patients in the safety population who have at least 1 assessment performed during the TEAE period. When a PCSA definition involves a change from baseline value, patients must also have a baseline value to be included in the summaries.

A listing of patients with at least 1 post-baseline PCSA will be provided and will display the patient's profile over time of all vital sign parameters. Individual data listings will include the following flags:

- Baseline values will be flagged "B".
- Parameter values reaching a PCSA limit will be flagged (+, or depending of the direction).

## 2.4.5.6 Analyses of electrocardiogram variables

Shift tables will be provided to present ECG status according to baseline status (Normal/Missing, Abnormal) for each treatment group during the TEAE period. Supportive listings of patients with abnormal ECG status at any post-baseline visit will be provided.

## 2.4.5.7 Analyses of physical examination variables

Shift tables will be provided to present physical examination findings by body system according to baseline status (Normal/Missing, Abnormal) for each treatment group during the TEAE period. Supportive listings of patients with abnormal findings at any post-baseline visit will be provided.

## 2.4.6 Analyses of pharmacokinetic variables

Plasma concentrations of sotagliflozin and its 3-O-glucuronide metabolite will be summarized by visit and nominal sampling time (pre-dose at Weeks 4, 18 and 26 and 3 hours post-dose at Week 26) in the PK population (see Section 2.3.3) in the sotagliflozin group, using descriptive statistics such as number, geometric mean, coefficient of variation, median, minimum and maximum. Individual plasma concentrations of sotagliflozin and its 3-O-glucuronide metabolite at nominal sampling times will also be listed.

#### 2.5 DATA HANDLING CONVENTIONS

#### 2.5.1 General conventions

The following formulas will be used for computation of parameters.

#### HbA1c

The formula to convert HbA1c from Diabetes Control and Complications Trial (DCCT) aligned value to International Federation of Clinical Chemistry and Laboratory Medicine (IFCC) standardized value is,

IFCC-HbA1c (mmol/mol) =  $[DCCT-HbA1c (\%) - 2.15] \times 10.929$ .

# Renal function formulas

The estimated GFR (mL/min/1.73 m<sup>2</sup>) will be calculated using the 4 variable Modification of Diet in Renal Disease (MDRD) formula:

Standard unit: eGFR (mL/min/1.73 m<sup>2</sup>) = 175 x [Serum Creatinine ( $\mu$ mol/L)/88.4] <sup>-1.154</sup> x Age (year) <sup>-0.203</sup> x 1.212 (if Black) x 0.742 (if female)

Conventional unit: eGFR (mL/min/1.73 m<sup>2</sup>) = 175 x Serum Creatinine (mg/dL)  $^{-1.154}$  x Age (year)  $^{-0.203}$  x 1.212 (if Black) x 0.742 (if Female)

#### Urine ACR

Standard unit: Urine ACR (mg/g) = Urine Albumin (mg/dL) / [Urine Creatinine (mmol/L)  $\times$  11.31]  $\times$  1000

Conventional unit: Urine ACR (mg/g) = Urine Albumin (mg/dL) / Urine Creatinine (mg/dL) x 1000

#### Urine GCR

Standard unit: Urine GCR = Urine Glucose (mmol/L) / Urine Creatinine (mmol/L)

Conventional unit: Urine GCR = Urine Glucose (mg/dL) / Urine Creatinine (mg/dL)

# Calculation of LDL-C

When TG is lower than or equal to 4.52 mmol/L (400 mg/dL), LDL-C is calculated using the Friedewald equation as:

- In standard unit (mmol/L), TC HDL-C TG/2.17.
- In conventional unit (mg/dL), TC HDL-C TG/5.

# 2.5.2 Data handling conventions for secondary efficacy variables

Scheduled measurements (see Section 2.5.4) of continuous efficacy variables collected during the study will be used in the analyses including those obtained after IMP discontinuation or introduction of rescue therapy. Continuous secondary efficacy endpoints will be analyzed with missing values imputed by retrieved dropout MI method (if there are at least 5 patients in each study treatment group who discontinued but have the endpoint) or washout MI method according to the criterion described in Section 2.4.4.1.

For the categorical secondary efficacy endpoints, data handling conventions are described in Section 2.4.4.2.

# 2.5.3 Missing data

For categorical variables, patients with missing data are not included in calculations of percentages unless otherwise specified. When relevant, the number of patients with missing data is presented.

Derived variables will be considered missing if any of the original variables required to calculate them are missing. For example, if either a baseline assessment or an endpoint assessment is missing for a particular patient, then change from baseline at endpoint will be missing. Depending

upon the assessment, analyses may not include all patients in the analysis population, because certain patients in the intended population may have missing data.

# Incomplete date of first administration of double-blind IMP

Date/time of first administration is the first non-missing start date/time of double-blind IMP completed in the e-CRF "First dose IMP" module.

For patients who are randomized and dispensed a double-blind treatment kit but who are lost to follow-up just after Visit 3 (eg. only the treatment kit number is reported in the e-CRF "Exposure - treatment period" module without any dose information), the date of first administration will be imputed using the date of randomization. When a patient is randomized but not exposed, "Not taken" should be ticked in the e-CRF "First dose IMP" module.

# Handling of computation of treatment duration if IMP end of treatment date is missing

For the calculation of the treatment duration, the date of the last dose of double-blind IMP is equal to the date of last administration reported on the e-CRF "Treatment status library" page. If this date is missing, the exposure duration should be left as missing.

The last dose administration should be clearly identified in the e-CRF and should not be approximated by the last returned package date.

# Handling of medication missing/partial dates

No imputation of medication start/end dates or times will be performed. If a medication date or time is missing or partially missing and it cannot be determined whether it was taken prior or concomitantly, it will be considered a prior, concomitant, and post-treatment medication.

#### Handling of adverse events/hypoglycemia with missing or partial date/time of onset

Missing or partial adverse event/hypoglycemia onset dates and times will be imputed so that if the partial adverse event/hypoglycemia onset date/time information does not indicate that the adverse event/hypoglycemia started prior to treatment or after the treatment-emergent adverse event period, the adverse event/hypoglycemia will be classified as treatment-emergent. No imputation of adverse event end dates/times will be performed. These data imputations are for categorization purpose only and will not be used in listings. No imputation is planned for date/time of adverse event resolution.

# Handling of adverse events/hypoglycemia when date and time of first IMP administration is missing

When the date and time of the first double-blind IMP administration is missing, the day of randomization should be considered as the start date of TEAE period (Section 2.1.4). The exposure duration should be kept as missing.

# Handling of adverse events/hypoglycemia when IMP end of treatment date is missing

For the purpose of defining TEAE period, the date of the last administration of double-blind IMP is equal to the date of the last administration reported on the e-CRF "Treatment Status Library" page.

If the date of last administration reported on the e-CRF "Treatment Status Library" page is

- Partially missing, it will be imputed with a date as late as possible before or on the date of last available information on e-CRF "Completion of End of Study/Follow-up".
- Completely missing, it will be imputed with the date of last available information on e-CRF "Completion of End of Study/Follow-up" page.

If the date of last available information on e-CRF "Completion of End of Study/Follow-up" page is

- Partially missing, it will be imputed with a date as late as possible.
- Completely missing, all adverse events occurred on or after the first administration of double-blind IMP will be considered as treatment emergent adverse events.

# Handling of missing assessment of relationship of adverse events to IMP (Capsule or Tablet)

If the assessment of the relationship to sotagliflozin or matching placebo (Tablet) is missing, the relationship to sotagliflozin or matching placebo (Tablet) has to be assumed. If the assessment of the relationship to empagliflozin or matching placebo (Capsule) is missing, the relationship to empagliflozin or matching placebo (Capsule) has to be assumed. The adverse event has to be considered as such in the frequency tables of possibly related adverse events, but no imputation should be done at the data level.

#### Handling of missing severity/grades of adverse events

If the severity/grade is missing for 1 of the treatment-emergent occurrences of an adverse event, the maximal severity on the remaining occurrences will be considered. If the severity is missing for all the occurrences, a "missing" category will be added in the summary table.

## Handling of potentially clinically significant abnormalities

If a patient has a missing baseline he will be grouped in the category "normal/missing at baseline."

For PCSAs with 2 conditions, one based on a change from baseline value or a normal range and the other on a threshold value, with the first condition being missing, the PCSA will be based only on the second condition.

For a PCSA defined on a threshold and/or a normal range, this PCSA will be derived using this threshold if the normal range is missing; eg, for eosinophils the PCSA is >0.5 GIGA/L or >ULN if ULN  $\geq$ 0.5 GIGA/L. When ULN is missing, the value 0.5 should be used.

Measurements flagged as invalid by the laboratory will not be summarized or taken into account in the computation of PCSA values.

#### Linked adverse events that worsened or became serious

An AE that worsened or became serious will have a separate record in the data from the original event record with an AE identification number that links the new record to the original record. An AE that worsened or became serious will be considered a new recurring AE in the summary of recurrent events or in the summary of events by time intervals.

# Handling of missing data for continuous efficacy endpoints

Please see Section 2.4.4.1 and Section 2.4.4.2.

# Handling of missing data for categorical efficacy endpoints

Please see Section 2.4.4.2.

## 2.5.4 Windows for time points /Measurements for analyses

The following steps will decide how the scheduled and/or unscheduled visits will be used in the analyses for efficacy variables and the by-visit summaries for safety variables (clinical laboratory data in Section 2.1.4.4 and vital signs in Section 2.1.4.5).

Step 1 A scheduled measurement will be used if it is available; otherwise, an unscheduled measurement (including the end of treatment/study visit for those prematurely discontinued) will be used if it happens to be on the same date as the date of the scheduled visit.

Step 2 After Step 1, if there are still no measurement for a given parameter at a scheduled visit, the analysis window below (Table 4) will be applied to re-allocate a post-baseline unscheduled measurement to a scheduled measurement.

Table 4 - Analyses window definition

| Scheduled visit post baseline | Targeted study day | Analysis window in study days |
|---|---|---|
| Main study | | |
| Week 4 (Visit 4) | 28 | 2 to 41 |
| Week 8 (Visit 5) | 56 | 42 to 69 |
| Week 12 (Visit 6) | 84 | 70 to 104 |
| Week 18 (Visit 7) | 126 | 105 to 153 |
| Week 26 (Visit 8) | 182 | ≥154 |
| ABPM substudy | | |
| Week 12 (Visit 6A) | 83 | 70 to 133 |

Version:3 Lexicon Pharmaceuticals Protocol No. EFC14867 **Date of Issue: 15-Nov-2019** Covance Study ID: 000000155204

| Scheduled visit post baseline | Targeted study day | Analysis window in study days |
|---|---|---|
| Main study | | |
| Week 26 (Visit 8A | 181 | ≥134 |

Study days are calculated from the day of first administration of double-blind IMP; the day of first administration of IMP (or the day of randomization if not exposed) is Day 1.

After applying the above time windows, if multiple assessments are associated to the same time point, the closest from the targeted study day will be used. In case of equality, the last measurement will be used. Re-allocated scheduled visits (ie, visit numbers) should be sequential if ordered by the date of measurement.

After Step 2, if there are still no measurement for a given parameter at a scheduled visit, data is considered missing for efficacy analyses, where multiple imputation would be applied as appropriately as described in Section 2.4.4.

# Reference day

The reference day for the calculation of extent of exposure, time to onset, and relative days will be the day of the first administration of double-blind IMP or the day of randomization if not exposed to double-blind IMP, denoted as Day 1.

# Baseline definition for efficacy/safety data

For the safety analyses, the baseline for a given parameter is defined as the last available measurement (or the average of all measurements for creatinine and eGFR), including unscheduled assessments, assessed prior to the first administration of double-blind IMP. For the efficacy analyses, the baseline for a given parameter is defined as the last available measurement (or the average of all measurements for creatinine and eGFR), including unscheduled assessments, assessed prior to the first administration of double-blind IMP or the last available value (or the average of all measurements for creatinine and eGFR) before randomization if not treated with double-blind IMP.

# Summary statistics by visit for continuous efficacy endpoints

Summary statistics (number, mean, SD, SE, minimum, median, maximum) of continuous efficacy endpoints (observed data and change from baseline) will be provided at scheduled visits as per protocol. Summaries showing data by visit will be presented according to the visit number (or re-allocated visit number, see Section 2.5.4) and labeled with the targeted approximate day/week.

# Last on-treatment value for laboratory variables and vital signs

The last on-treatment value is the final measurement assessed during the treatment epoch, regardless of the introduction of rescue therapy, including measurements at unscheduled visits. Please see details in Section 2.1.4 and Section 2.4.5.

# Display of safety data by visit (laboratory variables and vital signs)

Descriptive statistics (number, mean, SD, minimum, median, maximum) of quantitative laboratory variables and vital signs (observed data and change from baseline) during the TEAE period will be provided at scheduled visits. In addition, these summaries will also include a row for the 'last value on-treatment' to describe the last available on-treatment value (see above). Summaries showing data by visit will be presented according to the visit number (or re-allocated visit number, see Section 2.5.4) and labeled with the targeted approximate day/week.

As specified in the study protocol, laboratory data from scheduled visits are reported by central laboratories. The local results will not be used in the efficacy analyses or in the definition of baseline for both safety and efficacy analyses. In the safety analyses, for parameters with PCSA defined based on normal range, local results will only be used in the PCSA summary if they are accompanied by a local laboratory normal range. For parameters with PCSA not defined based on normal range, local results will be used in the PCSA summary as appropriately.

When a patient has more than 1 measurement from the central laboratory for the same laboratory parameter on the same date, the average of the measurements will be used. For the same laboratory parameter, if a patient has more than 1 measurement on different dates for the same scheduled visit, the value closest to the date of the visit will be used for the scheduled visit. When the values for the same scheduled visit are equidistant, the last value should be used for the scheduled visit. Similar rules will be applicable to a patient who has more than 1 set of measurements for the same vital sign parameter (ie, SBP, DBP, or HR) on the same date.

#### Time to event analysis

For time to event analysis/KM plot, time to event (eg, treatment discontinuation, rescue therapy, hypoglycemia, etc) is defined as the number of days from the date of the first administration of double-blind IMP (or the date of randomization if not exposed) to the start date of the first occurrence of the event during the 26-week double-blind treatment period.

Patients who did not experience any event during the 26-week double-blind treatment period are considered censored observations. For time to treatment discontinuation/rescue therapy, censoring date is the date of EOT. For time to severe or documented hypoglycemia, censoring date is the date of EOT+1 or the date of EOS, whichever is the earliest. Date of EOS will be used if the date of EOT is not available. Last contact date will be used if date of EOS is not available.

#### 2.5.5 Unscheduled visits

Unscheduled visit measurements of laboratory data, vital signs, and ECG will be used for computation of baseline, the last on-treatment value, PCSAs and the shift summaries for safety or efficacy. They will be included in the by-visit summaries if they are re-allocated to scheduled visit (see Section 2.5.4).

# 2.5.6 Pooling of centers for statistical analyses

Center will not be included in the statistical models for efficacy analyses. However, all centers within a country will be pooled, and country will be included as a fixed effect in a parametric statistical model (eg, ANCOVA etc) for primary and secondary efficacy endpoints. Countries with fewer than 5 randomized patients will be grouped, if patients from grouped countries are still fewer than 5, they will then be further grouped with the country with the lowest number of patients that is 5 or more.

#### 2.5.7 Statistical technical issues

None.

# 3 INTERIM ANALYSIS

No formal interim analysis for efficacy is planned for this study. The study will not be terminated early for excellent efficacy.

An independent Data Monitoring Committee (DMC) will be used to monitor and assess the safety of patients from this trial through periodic review of the accumulated safety data provided by an independent statistical group. Related details are provided in separate documents (DMC charter and DMC SAP).

# 4 DATABASE LOCK

The database lock was on 05Aug2019.

# 5 SOFTWARE DOCUMENTATION

All summaries and statistical analyses will be generated using SAS Version 9.2 or higher.

Lexicon Pharmaceuticals Protocol No. EFC14867

**Date of Issue: 15-Nov-2019** Covance Study ID: 000000155204

# **6 REFERENCES**

1. O'Brien E, Parati G, Stergiou G, Asmar R, Beilin L, Bilo G, et al. European Society of Hypertension position paper on ambulatory blood pressure monitoring. Journal of hypertension. 2013;31(9):1731-68.

# 7 LIST OF APPENDICES

| Appendix A | Ambulatory | blood | pressure | monitoring | substudy |
|-----------------|------------|-------|----------|------------|----------|
| i ippeliula 1 i | Impulatory | UIUUU | prossure | momornia | substuay |

Appendix B ABPM substudy efficacy variable derivation

Appendix C List of PTs for select EOSIs (MedDRA v22.0)

Appendix D Potentially clinically significant abnormalities criteria

Appendix E Summary of statistical analyses

Appendix F Study Flow Chart

# Appendix A Ambulatory blood pressure monitoring substudy

# **Background**

A Phase 2 trial of sotagliflozin (LX4211.1-202) provided evidence that sotagliflozin reduced both SBP and DBP in patients with elevated SBP and DBP at baseline but not normotensive patients. In this substudy of approximately 180 patients, patients with similar Baseline BP distribution as the full study population (ie, equal numbers of patients with SBP <130 mmHg or ≥130 mmHg) will have ABPM assessed for 24 hours via ambulatory BP monitoring technology at baseline, Week 12, and Week 26 to provide a more systematic assessment of the SBP and DBP lowering efficacy of sotagliflozin.

# **Substudy procedures**

At the preselected study sites participating in the ABPM substudy, patients must consent to be a part of the substudy to participate in the main study until the planned number of patients for substudy has been achieved.

At Visit 1, patients will be provided with information on the ABPM substudy and separate written consent will be taken before ABPM substudy-specific procedures are performed. Patients who work a night (third) shift (defined as 11:00 PM [23:00] to 7:00 AM [07:00]) will be excluded from the ABPM substudy.

Patients in the ABPM substudy will have 3 additional visits to the site for placement of the ABPM device. These will be Visits 3A, 6A, and 8A. Visit 3A will occur at Week -1, 1 week before the Randomization Visit. Visit 6A, and Visit 8A will occur the day before Visit 6 (Week 12) and Visit 8 (Week 26). Patients do not need to be fasting at these 3 visits.

Patients who discontinued the Investigational Medicinal Product (IMP) during the study before the visit for ABPM will not continue in the ABPM substudy post-IMP discontinuation. Patients who receive rescue therapy but remain on IMP will continue on the ABPM substudy as planned.

On the 3 visit days (Visits 3A, 6A, and 8A) each recording will start in the morning, preferably between 08:00 and 10:00 immediately after the administration of study medication, and will end after at least 24 hours of recording on the following day.

- Investigator and/or designee will help patients wear the ambulant BP monitor and the appropriate BP cuff (depending on the patient's arm size) on the nondominant upper arm.
- Patients should be aware that the device will automatically inflate the cuff and measure the BP every 20 minutes during the day-time (08:00 and 21:59) and every 30 minutes during the sleeping time (22:00 and 07:59) over a 24-hour period.
- During the ABPM period, patients should continue their daily activities and concomitant medications, but avoid activities that may interfere with functioning of the device such as vigorous exercise, bathing, or taking a shower.

- When the cuff starts to inflate, the patient should remain still and avoid arm movement.
- Patients will record the time of sleep and any unusual events or poor sleep quality during the ABPM recording period in their study diary.
- Patients will be instructed to remove the BP device after 24-hour wearing the ABPM device:
  - Once the ABPM device has been placed at Visit 3A, patients will be instructed to remove it 24 hours later and return it to the site by mail in appropriate packaging provided by the site?
  - Twenty-four hours after Visits 6A and 8A, patients will return to the site in a fasting state at Visits 6 and 8, respectively, and the device will be removed at the site.

All ABPM data will be reviewed following return of the device to ensure quality of the recording. Patients with ABPM data not of sufficient quality will be asked to repeat the process as soon as possible. Patients with ABPM data not of sufficient quality at Visit 3A should not be randomized until the Baseline ABPM recording has been repeated, and the Randomization Visit (Visit 3) will be postponed correspondingly.

# **Sub-study objectives**

The objective of the ABPM substudy is to compare the effect of sotagliflozin, empagliflozin and placebo for a subset of patients based on:

- 24-hour average SBP and DBP.
- Average adjusted awake time BP as measured by SBP and DBP with adjustment based on actigraphy.
- Average adjusted sleeping time BP as measured by SBP and DBP with adjustment based on actigraphy.

# **Sub-study endpoints**

The ABPM endpoints are changes from Baseline to Week 12 and Week 26 for all patients participating substudy, patients with baseline 24-hour average SBP≥130 mmHg and patients with baseline 24-hour average SBP<130 mmHg in:

- 24-hour average SBP and DBP.
- Average adjusted awake time BP as measured by SBP and DBP with adjustment based on actigraphy.

Date of Issue: 15-Nov-2019 Lexicon Pharmaceuticals Protocol No. EFC14867 Covance Study ID: 000000155204

Average adjusted sleeping time BP as measured by SBP and DBP with adjustment based on actigraphy.

# Statistical analyses

The quality of a visit recording will be considered insufficient if the visit recording does not meet the criteria below (1):

- 1. Visit recording does not contain  $\ge 17$  nonconsecutive hours of data where each hour has at least one valid BP measurement.
- 2. Visit recording has <44 total measurements.

Analyses of ABPM substudy efficacy endpoints will be performed on the ABPM population using all assessment collected up to Week 26. All ABPM substudy efficacy endpoints will be summarized by descriptive statistics by scheduled visits (Baseline (Visit 3A, Week -1), Visit 6A (Week 12), and Visit 8A (Week 26)). The descriptive statistics will include number, mean, standard deviation, Q1, Q3, minimum, maximum. In addition, analyses will be done for those patients with baseline Mean 24-hour SBP ≥130 mmHg and those patients with baseline Mean 24-hour SBP <130 mmHg separately.

# Appendix B ABPM substudy efficacy variable derivation

| All following derivation of the | efficacy variables for | ABPM substudy will be performed and |
|---|---|---|
| provided by vendor (special | alized in ABPM device | ce) by using validated software |
| | and following | Project Requirement Specifications as |
| follows: | | |

All ABPM substudy efficacy measurements will be recorded by validated ABPM Ambulo 2400 device. The device's inflation plan is set up to collect patient's BP measurements every 20 minutes during 8:00-21:59 and every 30 minutes during 22:00 -7:59 over at least 24-hour time interval. The device will start recording patient's blood pressure after its inflation is initiated, which composes a patient's visit recording. All individual measurements will be analyzed by and be assigned a status of successful included, successful excluded manual inflations, error or event.

Successful excluded measurements are valid device log entries related to manual device initiation of inflation by the patient and will be excluded from analysis. Error measurements are any attempted inflation that results in a 0 value for one of the four values the device captures: systolic, diastolic, mean atrial pressure, or pulse pressure. Examples of errors are "cuff leak," device error, movement error, etc. These errors could be the result of a hole in the hose or patient movement (during inflation or deflation of the cuff). Events refer to non-inflation events which appear in the data with 0 values for systolic, diastolic, mean atrial pressure, and pulse pressure. Examples of these events are USB disconnect, sequence trigger, and power on reset. Usually, occurrence of events will not impact the quality of the recording. Both events and errors are excluded from analysis. Successful included measurements are device log entries during the time interval after device automatic initiation based on the inflation plan (daytime, nighttime, or 24-hour period) that are neither successful excluded manual inflation plan, error, nor event. The successful included measurement captured systolic, diastolic, mean atrial pressure, and pulse pressure.

The quality of each recording at each visit will be considered Not Good Quality and not acceptable for analysis if the visit recording meets the criteria below:

- 1. Visit Recording does not contain greater than or equal to 17 non-consecutive hours of data where each hour has at least one valid BP measurement.
- 2. Visit Recording has less than 44 total measurements.

A valid measurement is a measurement having non-missing values for systolic, diastolic, pulse pressure and mean arterial pressure (MAP). will analyze the recording from the first valid inflation (after device initiated) up to 24 hours thereafter to determine the quality of the recording. If the quality of the visit recording is of Not Good Quality, the efficacy variable of the patient at that visit will be considered as missing value. Otherwise, the efficacy variable of the patient at the visit will be calculated as follow:

Summing over all successful included systolic/diastolic measurements collected during the time interval (24-hour, actigraphy reported sleep time or actigraphy reported wake time), then divide the total by number of successful included measurements.

#### **Statistical Analysis Plan**

**Version:3**Lexicon Pharmaceuticals Protocol No. EFC14867

**Date of Issue: 15-Nov-2019**Covance Study ID: 000000155204

The actigraphy can detect the patient's sleep or wake time based on the patient's activity intensity. If the patient has interruptive sleep periods, the actigraphy will report the first inactivity period of the patient as the patient's sleep time. Wake time will be the time outside the sleep interval. Each patient will only have one sleep time and one wake time reported by the device.

# Appendix C List of PTs for select EOSIs (MedDRA v22.0)

| EOSI | Preferred | Preferred Term |
|---|---|---|
| | Term Code | |
| Genital Mycotic Infections | 10004074 | Balanitis candida |
| Genital Mycotic Infections | 10018143 | Genital candidiasis |
| Genital Mycotic Infections | 10047784 | Vulvovaginal candidiasis |
| Genital Mycotic Infections | 10061180 | Genital infection fungal |
| Genital Mycotic Infections | 10064899 | Vulvovaginal mycotic infection |
| Genital Mycotic Infections | 10065582 | Urogenital infection fungal |
| Genital Mycotic Infections | 10071209 | Candida cervicitis |
| Genital Mycotic Infections | 10079521 | Fungal balanitis |
| Urinary tract infections | 10011781 | Cystitis |
| Urinary tract infections | 10011790 | Cystitis escherichia |
| Urinary tract infections | 10011797 | Cystitis klebsiella |
| Urinary tract infections | 10011799 | Cystitis pseudomonal |
| Urinary tract infections | 10017525 | Fungal cystitis |
| Urinary tract infections | 10018185 | Genitourinary chlamydia infection |
| Urinary tract infections | 10023424 | Kidney infection |
| Urinary tract infections | 10037584 | Pyelitis |
| Urinary tract infections | 10037596 | Pyelonephritis |
| Urinary tract infections | 10037597 | Pyelonephritis acute |
| Urinary tract infections | 10037601 | Pyelonephritis chronic |
| Urinary tract infections | 10037603 | Pyelonephritis mycoplasmal |
| Urinary tract infections | 10037653 | Pyonephrosis |
| Urinary tract infections | 10038351 | Renal abscess |
| Urinary tract infections | 10044828 | Tuberculosis of genitourinary system |
| Urinary tract infections | 10046424 | Urethral abscess |
| Urinary tract infections | 10046480 | Urethritis |
| Urinary tract infections | 10046482 | Urethritis chlamydial |
| Urinary tract infections | 10046483 | Urethritis gonococcal |
| Urinary tract infections | 10046490 | Urethritis ureaplasmal |
| Urinary tract infections | 10046571 | Urinary tract infection |
| Urinary tract infections | 10046572 | Urinary tract infection enterococcal |
| Urinary tract infections | 10046704 | Urogenital trichomoniasis |
| Urinary tract infections | 10048302 | Tubulointerstitial nephritis |
| Urinary tract infections | 10048709 | Urosepsis |
| Urinary tract infections | 10048709 | Cystitis glandularis |
| Urinary tract infections | 10048837 | Urinary tract infection fungal |
| Urinary tract infections | 10049039 | Pyelocystitis |
| Urinary tract infections | | Ureteritis |
| • | 10051250 | |
| Urinary tract infections | 10051350 | Cytomegalovirus urinary tract infection |
| Urinary tract infections | 10051959 | Urinary bladder abscess |
| Urinary tract infections | 10052238 | Escherichia urinary tract infection |
| Urinary tract infections | 10054088 | Urinary tract infection bacterial |
| Urinary tract infections | 10056351 | Emphysematous cystitis |
| Urinary tract infections | 10058523 | Bladder candidiasis |
| Urinary tract infections | 10058596 | Renal cyst infection |
| Version:3 Lexicon Pharmaceuticals Protocol No. EFC14867 | | Date of Issue: 15-Nov-2019<br>Covance Study ID: 000000155204 | |
|---|---|---|--|
| Urinary tract infections | 10059517 | Bacterial pyelonephritis | |
| Urinary tract infections | 10061181 | Genitourinary tract gonococcal infection | |
| Urinary tract infections | 10061182 | Genitourinary tract infection | |
| Urinary tract infections | 10061395 | Ureter abscess | |
| Urinary tract infections | 10062279 | Urinary tract infection pseudomonal | |
| Urinary tract infections | 10062280 | Urinary tract infection staphylococcal | |
| Urinary tract infections | 10064825 | Urinary tract infection viral | |
| Urinary tract infections | 10064921 | Urinary tract inflammation | |
| Urinary tract infections | 10065197 | Cystitis viral | |
| Urinary tract infections | 10065198 | Cystitis bacterial | |
| Urinary tract infections | 10065199 | Cystitis helminthic | |
| Urinary tract infections | 10065213 | Pyelonephritis viral | |
| Urinary tract infections | 10065214 | Pyelonephritis fungal | |
| Urinary tract infections | 10065582 | Urogenital infection fungal | |
| Urinary tract infections | 10065583 | Urogenital infection bacterial | |
| Urinary tract infections | 10066757 | Urinary tract abscess | |
| Urinary tract infections | 10068822 | Emphysematous pyelonephritis | |
| Urinary tract infections | 10070300 | Streptococcal urinary tract infection | |
| Urinary tract infections | 10074409 | Escherichia pyelonephritis | |
| Urinary tract infections | 10075063 | Urethritis mycoplasmal | |
| Urinary tract infections | 10078665 | Bacterial urethritis | |
| Urinary tract infections | 10081163 | Fungal urethritis | |
| Urinary tract infections | 10081262 | Candida urethritis | |
| Urinary tract infections | 10082040 | Nephritis bacterial | |
| Volume depletion | 10005697 | Blood osmolarity increased | |
| Volume depletion | 10005731 | Blood pressure ambulatory decreased | |
| Volume depletion | 10005734 | Blood pressure decreased | |
| Volume depletion | 10005737 | Blood pressure diastolic decreased | |
| Volume depletion | 10005748 | Blood pressure immeasurable | |
| Volume depletion | 10005758 | Blood pressure systolic decreased | |
| Volume depletion | 10005761 | Blood pressure systolic inspiratory decreased | |
| Volume depletion | 10007979 | Central venous pressure decreased | |
| Volume depletion | 10009192 | Circulatory collapse | |
| Volume depletion | 10012174 | Dehydration | |
| Volume depletion | 10013578 | Dizziness postural | |
| Volume depletion | 10021097 | Hypotension | |
| Volume depletion | 10021137 | Hypovolaemia | |
| Volume depletion | 10021138 | Hypovolaemic shock | |
| Volume depletion | 10026983 | Mean arterial pressure decreased | |
| Volume depletion | 10031127 | Orthostatic hypotension | |
| Volume depletion | 10036653 | Presyncope | |
| Volume depletion | 10037327 | Pulmonary arterial wedge pressure decreased | |
| Volume depletion | 10042772 | Syncope | |
| Volume depletion | 10046640 | Urine flow decreased | |
| Volume depletion | 10047235 | Venous pressure decreased | |
| Volume depletion | 10047239 | Venous pressure jugular decreased | |

| Version:3 Lexicon Pharmaceuticals Protocol No. EFC14867 | | Date of Issue: 15-Nov-2019<br>Covance Study ID: 000000155204 |
|---|---|---|
| Volume depletion | 10047689 | Volume blood decreased |
| Volume depletion | 10050760 | Blood urea nitrogen/creatinine ratio increased |
| Volume depletion | 10050905 | Decreased ventricular preload |
| Volume depletion | 10053356 | Blood pressure orthostatic decreased |
| Volume depletion | 10059895 | Urine output decreased |
| Volume depletion | 10060089 | Left ventricular end-diastolic pressure decreased |
| Volume depletion | 10060231 | Pulmonary arterial pressure decreased |
| Volume depletion | 10063080 | Postural orthostatic tachycardia syndrome |
| Volume depletion | 10063927 | Orthostatic intolerance |
| Volume depletion | 10066077 | Diastolic hypotension |
| Volume depletion | 10069431 | Orthostatic heart rate response increased |
| Volume depletion | 10069583 | Pulse volume decreased |
| Volume depletion | 10072370 | Prerenal failure |
| Pancreatitis | 10033625 | Pancreatic haemorrhage |
| Pancreatitis | 10033635 | Pancreatic pseudocyst |
| Pancreatitis | 10033636 | Pancreatic pseudocyst drainage |
| Pancreatitis | 10033645 | Pancreatitis |
| Pancreatitis | 10033647 | Pancreatitis acute |
| Pancreatitis | 10033649 | Pancreatitis chronic |
| Pancreatitis | 10033650 | Pancreatitis haemorrhagic |
| Pancreatitis | 10033654 | Pancreatitis necrotising |
| Pancreatitis | 10033657 | Pancreatitis relapsing |
| Pancreatitis | 10048984 | Pancreatic abscess |
| Pancreatitis Pancreatitis | 10052400<br>10056277 | Oedematous pancreatitis |
| Pancreatitis | 10056277 | Pancreatorenal syndrome Pancreatic phlegmon |
| Pancreatitis | 10056976 | Hereditary pancreatitis |
| Pancreatitis | 10056977 | Alcoholic pancreatitis |
| Pancreatitis | 10058096 | Pancreatic necrosis |
| Pancreatitis | 10065189 | Pancreatitis helminthic |
| Pancreatitis | 10066127 | Ischaemic pancreatitis |
| Pancreatitis | 10069002 | Autoimmune pancreatitis |
| Pancreatitis | 10074894 | Traumatic pancreatitis |
| Pancreatitis | 10076058 | Haemorrhagic necrotic pancreatitis |
| Venous thrombotic events | 10003192 | Arteriovenous fistula thrombosis |
| Venous thrombotic events | 10003880 | Axillary vein thrombosis |
| Venous thrombotic events | 10006537 | Budd-Chiari syndrome |
| Venous thrombotic events | 10007830 | Cavernous sinus thrombosis |
| Venous thrombotic events | 10008138 | Cerebral venous thrombosis |
| Venous thrombotic events | 10014522 | Embolism venous |
| Venous thrombotic events | 10019713 | Hepatic vein thrombosis |
| Venous thrombotic events | 10023237 | Jugular vein thrombosis |
| Venous thrombotic events | 10027402 | Mesenteric vein thrombosis |
| Venous thrombotic events | 10034272 | Pelvic venous thrombosis |
| Venous thrombotic events | 10034324 | Penile vein thrombosis |
| Venous thrombotic events | 10036206 | Portal vein thrombosis |

| Version:3 | | Date of Issue: 15-Nov-2019 |
|---|---|---|
| Lexicon Pharmaceuticals Protocol N | | Covance Study ID: 000000155204 |
| Venous thrombotic events | 10037377 | Pulmonary embolism |
| Venous thrombotic events | 10037421 | Pulmonary microemboli |
| Venous thrombotic events | 10037437 | Pulmonary thrombosis |
| Venous thrombotic events | 10037459 | Pulmonary venous thrombosis |
| Venous thrombotic events | 10038547 | Renal vein embolism |
| Venous thrombotic events | 10038548 | Renal vein thrombosis |
| Venous thrombotic events | 10038908 | Retinal vein thrombosis |
| Venous thrombotic events | 10041659 | Splenic vein thrombosis |
| Venous thrombotic events | 10042567 | Superior sagittal sinus thrombosis |
| Venous thrombotic events | 10043570 | Thrombophlebitis |
| Venous thrombotic events | 10043581 | Thrombophlebitis migrans |
| Venous thrombotic events | 10043595 | Thrombophlebitis superficial |
| Venous thrombotic events | 10043605 | Thrombosed varicose vein |
| Venous thrombotic events | 10044457 | Transverse sinus thrombosis |
| Venous thrombotic events | 10047193 | Vena cava embolism |
| Venous thrombotic events | 10047195 | Vena cava thrombosis |
| Venous thrombotic events | 10047249 | Venous thrombosis |
| Venous thrombotic events | 10048591 | Post thrombotic syndrome |
| Venous thrombotic events | 10049446 | Subclavian vein thrombosis |
| Venous thrombotic events | 10050216 | Paget-Schroetter syndrome |
| Venous thrombotic events | 10050902 | Postoperative thrombosis |
| Venous thrombotic events | 10051055 | Deep vein thrombosis |
| Venous thrombotic events | 10053182 | Arteriovenous graft thrombosis |
| Venous thrombotic events | 10061251 | Intracranial venous sinus thrombosis |
| Venous thrombotic events | 10061408 | Venous thrombosis limb |
| Venous thrombotic events | 10063363 | Brachiocephalic vein thrombosis |
| Venous thrombotic events | 10063909 | Post procedural pulmonary embolism |
| Venous thrombotic events | 10066881 | Deep vein thrombosis postoperative |
| Venous thrombotic events | 10067270 | Thrombosis corpora cavernosa |
| Venous thrombotic events | 10069909 | Metastatic pulmonary embolism |
| Venous thrombotic events | 10072059 | Ovarian vein thrombosis |
| Venous thrombotic events | 10074349 | Ophthalmic vein thrombosis |
| Venous thrombotic events | 10077623 | Portosplenomesenteric venous thrombosis |
| Venous thrombotic events | 10077829 | Visceral venous thrombosis |
| Venous thrombotic events | 10078810 | Hepatic vein embolism |
| Thyroid cancer | 10002240 | Anaplastic thyroid cancer |
| Thyroid cancer | 10016935 | Follicular thyroid cancer |
| Thyroid cancer | 10027105 | Medullary thyroid cancer |
| Thyroid cancer | 10033701 | Papillary thyroid cancer |
| Thyroid cancer | 10043744 | Thyroid neoplasm |
| Thyroid cancer | 10055107 | Thyroid cancer metastatic |
| Thyroid cancer | 10066136 | Huerthle cell carcinoma |
| Thyroid cancer | 10066474 | Thyroid cancer |
| Thyroid cancer | 10070567 | Thyroid cancer stage 0 |
| Thyroid cancer | 10071027 | Thyroid cancer stage I |
| Thyroid cancer | 10071028 | Thyroid cancer stage II |

| Version:3<br>Lexicon Pharmaceuticals Protocol No. EFC14867 | | Date of Issue: 15-Nov-2019<br>Covance Study ID: 000000155204 |
|---|---|---|
| Thyroid cancer | 10071029 | Thyroid cancer stage III |
| Thyroid cancer | 10071030 | Thyroid cancer stage IV |
| Thyroid cancer | 10072162 | Thyroid cancer recurrent |
| Thyroid cancer | 10072613 | Thyroid B-cell lymphoma |
| Thyroid cancer | 10073153 | Familial medullary thyroid cancer |
| Thyroid cancer | 10076603 | Poorly differentiated thyroid carcinoma |
| Renal cell cancer | 10038389 | Renal cancer |
| Renal cell cancer | 10038390 | Renal cancer recurrent |
| Renal cell cancer | 10038391 | Renal cancer stage I |
| Renal cell cancer | 10038392 | Renal cancer stage II |
| Renal cell cancer | 10038393 | Renal cancer stage III |
| Renal cell cancer | 10038394 | Renal cancer stage IV |
| Renal cell cancer | 10038410 | Renal cell carcinoma recurrent |
| Renal cell cancer | 10038411 | Renal cell carcinoma stage I |
| Renal cell cancer | 10038412 | Renal cell carcinoma stage II |
| Renal cell cancer | 10038413 | Renal cell carcinoma stage III |
| Renal cell cancer | 10038414 | Renal cell carcinoma stage IV |
| Renal cell cancer | 10050018 | Renal cancer metastatic |
| Renal cell cancer | 10050513 | Metastatic renal cell carcinoma |
| Renal cell cancer | 10061482 | Renal neoplasm |
| Renal cell cancer | 10067944 | Hereditary leiomyomatosis renal cell carcinoma |
| Renal cell cancer | 10067946 | Renal cell carcinoma |
| Renal cell cancer | 10073251 | Clear cell renal cell carcinoma |
| Renal cell cancer | 10078493 | Papillary renal cell carcinoma |
| Pancreatic cancer | 10018404 | Glucagonoma |
| Pancreatic cancer | 10022498 | Insulinoma |
| Pancreatic cancer | 10025997 | Malignant neoplasm of islets of Langerhans |
| Pancreatic cancer | 10029341 | Neurotensinoma |
| Pancreatic cancer | 10033609 | Pancreatic carcinoma |
| Pancreatic cancer | 10033610 | Pancreatic carcinoma metastatic |
| Pancreatic cancer | 10033613 | Pancreatic carcinoma recurrent |
| Pancreatic cancer | 10041329 | Somatostatinoma |
| Pancreatic cancer | 10047430 | Vipoma |
| Pancreatic cancer | 10051709 | Gastrinoma malignant |
| Pancreatic cancer | 10052747 | Adenocarcinoma pancreas |
| Pancreatic cancer | 10055006 | Pancreatic sarcoma |
| Pancreatic cancer | 10055007 | Carcinoid tumour of the pancreas |
| Pancreatic cancer | 10059320 | Pancreatic carcinoma stage 0 |
| Pancreatic cancer | 10059321 | Pancreatic carcinoma stage I |
| Pancreatic cancer | 10059322 | Pancreatic carcinoma stage II |
| Pancreatic cancer | 10059323 | Pancreatic carcinoma stage III |
| Pancreatic cancer | 10059326 | Pancreatic carcinoma stage IV |
| Pancreatic cancer | 10061902 | Pancreatic neoplasm |
| Pancreatic cancer | 10067517 | Pancreatic neuroendocrine tumour |
| Pancreatic cancer | 10068909 | Pancreatic neuroendocrine tumour metastatic |
| Pancreatic cancer | 10069345 | Solid pseudopapillary tumour of the pancreas |

| <br>Date of Issue: 15-Nov-2019 |
|--------------------------------|
| Covance Study ID: 000000155204 |

| Lexicon Pharmaceuticals Protocol No. EFC14867 | | Covance Study ID: 000000155204 |
|---|---|---|
| Pancreatic cancer | 10073363 | Acinar cell carcinoma of pancreas |
| Pancreatic cancer | 10073364 | Ductal adenocarcinoma of pancreas |
| Pancreatic cancer | 10073365 | Intraductal papillary-mucinous carcinoma of |
| | | pancreas |
| Pancreatic cancer | 10073367 | Pancreatoblastoma |
| Bladder cancer | 10004986 | Bladder adenocarcinoma recurrent |
| Bladder cancer | 10004987 | Bladder adenocarcinoma stage 0 |
| Bladder cancer | 10004988 | Bladder adenocarcinoma stage I |
| Bladder cancer | 10004989 | Bladder adenocarcinoma stage II |
| Bladder cancer | 10004990 | Bladder adenocarcinoma stage III |
| Bladder cancer | 10004991 | Bladder adenocarcinoma stage IV |
| Bladder cancer | 10004992 | Bladder adenocarcinoma stage unspecified |
| Bladder cancer | 10005003 | Bladder cancer |
| Bladder cancer | 10005005 | Bladder cancer recurrent |
| Bladder cancer | 10005006 | Bladder cancer stage 0, with cancer in situ |
| Bladder cancer | 10005007 | Bladder cancer stage 0, without cancer in situ |
| Bladder cancer | 10005008 | Bladder cancer stage I, with cancer in situ |
| Bladder cancer | 10005009 | Bladder cancer stage I, without cancer in situ |
| Bladder cancer | 10005010 | Bladder cancer stage II |
| Bladder cancer | 10005011 | Bladder cancer stage III |
| Bladder cancer | 10005012 | Bladder cancer stage IV |
| Bladder cancer | 10005056 | Bladder neoplasm |
| Bladder cancer | 10005075 | Bladder squamous cell carcinoma recurrent |
| Bladder cancer | 10005076 | Bladder squamous cell carcinoma stage 0 |
| Bladder cancer | 10005077 | Bladder squamous cell carcinoma stage I |
| Bladder cancer | 10005078 | Bladder squamous cell carcinoma stage II |
| Bladder cancer | 10005079 | Bladder squamous cell carcinoma stage III |
| Bladder cancer | 10005080 | Bladder squamous cell carcinoma stage IV |
| Bladder cancer | 10005081 | Bladder squamous cell carcinoma stage unspecified |
| Bladder cancer | 10005084 | Bladder transitional cell carcinoma |
| Bladder cancer | 10051690 | Urinary bladder sarcoma |
| Bladder cancer | 10057352 | Metastatic carcinoma of the bladder |
| Bladder cancer | 10066749 | Bladder transitional cell carcinoma stage 0 |
| Bladder cancer | 10066750 | Bladder transitional cell carcinoma recurrent |
| Bladder cancer | 10066751 | Bladder transitional cell carcinoma stage I |
| Bladder cancer | 10066752 | Bladder transitional cell carcinoma stage IV |
| Bladder cancer | 10066753 | Bladder transitional cell carcinoma stage II |
| Bladder cancer | 10066754 | Bladder transitional cell carcinoma stage III |
| Bladder cancer | 10071664 | Bladder transitional cell carcinoma metastatic |
| Bladder cancer | 10078341 | Neuroendocrine carcinoma of the bladder |
| Potentially leading to amputation | 10003084 | Areflexia |
| Potentially leading to amputation | 10003178 | Arterial thrombosis |
| Potentially leading to amputation | 10003210 | Arteriosclerosis |
| Potentially leading to amputation | 10003222 | Arteriosclerotic gangrene |
| Potentially leading to amputation | 10006784 | Burning sensation |

| Version:3 | | Date of Issue: 15-Nov-2019 |
|---|---|---|
| Lexicon Pharmaceuticals Protocol No. E | FC14867 | Covance Study ID: 000000155204 |
| Potentially leading to amputation | 10007904 | Cellulitis enterococcal |
| Potentially leading to amputation | 10007905 | Cellulitis gangrenous |
| Potentially leading to amputation | 10007921 | Cellulitis staphylococcal |
| Potentially leading to amputation | 10007922 | Cellulitis streptococcal |
| Potentially leading to amputation | 10012174 | Dehydration |
| Potentially leading to amputation | 10012665 | Diabetic gangrene |
| Potentially leading to amputation | 10012679 | Diabetic neuropathic ulcer |
| Potentially leading to amputation | 10012680 | Diabetic neuropathy |
| Potentially leading to amputation | 10017711 | Gangrene |
| Potentially leading to amputation | 10020937 | Hypoaesthesia |
| Potentially leading to amputation | 10021137 | Hypovolaemia |
| Potentially leading to amputation | 10021519 | Impaired healing |
| Potentially leading to amputation | 10021784 | Infected skin ulcer |
| Potentially leading to amputation | 10022562 | Intermittent claudication |
| Potentially leading to amputation | 10024774 | Localised infection |
| Potentially leading to amputation | 10028862 | Necrosis ischaemic |
| Potentially leading to amputation | 10029331 | Neuropathy peripheral |
| Potentially leading to amputation | 10031149 | Osteitis |
| Potentially leading to amputation | 10031252 | Osteomyelitis |
| Potentially leading to amputation | 10031253 | Osteomyelitis acute |
| Potentially leading to amputation | 10031256 | Osteomyelitis chronic |
| Potentially leading to amputation | 10031262 | Osteomyelitis salmonella |
| Potentially leading to amputation | 10031264 | Osteonecrosis |
| Potentially leading to amputation | 10033775 | Paraesthesia |
| Potentially leading to amputation | 10034568 | Peripheral coldness |
| Potentially leading to amputation | 10034576 | Peripheral ischaemia |
| Potentially leading to amputation | 10034620 | Peripheral sensory neuropathy |
| Potentially leading to amputation | 10034636 | Peripheral vascular disorder |
| Potentially leading to amputation | 10036155 | Poor peripheral circulation |
| Potentially leading to amputation | 10036410 | Postoperative wound infection |
| Potentially leading to amputation | 10040026 | Sensory disturbance |
| Potentially leading to amputation | 10040840 | Skin erosion |
| Potentially leading to amputation | 10040872 | Skin infection |
| Potentially leading to amputation | 10040943 | Skin ulcer |
| Potentially leading to amputation | 10042343 | Subcutaneous abscess |
| Potentially leading to amputation | 10043607 | Thrombosis |
| Potentially leading to amputation | 10048031 | Wound dehiscence |
| Potentially leading to amputation | 10048038 | Wound infection |
| Potentially leading to amputation | 10049927 | Dry gangrene |
| Potentially leading to amputation | 10050473 | Abscess limb |
| Potentially leading to amputation | 10050502 | Neuropathic ulcer |
| Potentially leading to amputation | 10051548 | Burn infection |
| Potentially leading to amputation | 10052428 | Wound |
| Potentially leading to amputation | 10052949 | Arterial therapeutic procedure |
| Potentially leading to amputation | 10053692 | Wound complication |
| Potentially leading to amputation | 10053716 | Wound necrosis |
| Potentially leading to amputation | 10054044 | Diabetic microangiopathy |
| Potentially leading to amputation | 10056340 | Diabetic ulcer |
| Potentially leading to amputation | 10056418 | Arterial bypass operation |

| Lexicon Pharmaceuticals Protocol No. E | EFC14867 | Covance Study ID: 000000155204 |
|---|---|---|
| Potentially leading to amputation | 10056673 | Peripheral sensorimotor neuropathy |
| Potentially leading to amputation | 10057518 | Peripheral artery angioplasty |
| Potentially leading to amputation | 10057525 | Peripheral artery occlusion |
| Potentially leading to amputation | 10058041 | Wound sepsis |
| Potentially leading to amputation | 10058042 | Wound abscess |
| Potentially leading to amputation | 10059245 | Angiopathy |
| Potentially leading to amputation | 10059385 | Extremity necrosis |
| Potentially leading to amputation | 10059442 | Wound infection staphylococcal |
| Potentially leading to amputation | 10059444 | Wound infection pseudomonas |
| Potentially leading to amputation | 10060734 | Diabetic foot |
| Potentially leading to amputation | 10060803 | Diabetic foot infection |
| Potentially leading to amputation | 10060963 | Arterial disorder |
| Potentially leading to amputation | 10060965 | Arterial stenosis |
| Potentially leading to amputation | 10061627 | Amputation |
| Potentially leading to amputation | 10061655 | Arterial graft |
| Potentially leading to amputation | 10061657 | Arterial stent insertion |
| Potentially leading to amputation | 10061666 | Autonomic neuropathy |
| Potentially leading to amputation | 10061815 | Diabetic vascular disorder |
| Potentially leading to amputation | 10062198 | Microangiopathy |
| Potentially leading to amputation | 10062255 | Soft tissue infection |
| Potentially leading to amputation | 10062585 | Peripheral arterial occlusive disease |
| Potentially leading to amputation | 10062599 | Arterial occlusive disease |
| Potentially leading to amputation | 10062610 | Ischaemic limb pain |
| Potentially leading to amputation | 10062932 | Wound treatment |
| Potentially leading to amputation | 10064250 | Staphylococcal osteomyelitis |
| Potentially leading to amputation | 10064601 | Iliac artery occlusion |
| Potentially leading to amputation | 10065237 | Osteomyelitis bacterial |
| Potentially leading to amputation | 10065239 | Osteomyelitis fungal |
| Potentially leading to amputation | 10065240 | Wound infection bacterial |
| Potentially leading to amputation | 10065242 | Wound infection fungal |
| Potentially leading to amputation | 10068653 | Bone abscess |
| Potentially leading to amputation | 10069379 | Peripheral arterial reocclusion |
| Potentially leading to amputation | 10072170 | Skin wound |
| Potentially leading to amputation | 10072557 | Peripheral artery restenosis |
| Potentially leading to amputation | 10072560 | Peripheral endarterectomy |
| Potentially leading to amputation | 10072561 | Peripheral artery bypass |
| Potentially leading to amputation | 10072562 | Peripheral artery stent insertion |
| Potentially leading to amputation | 10072563 | Peripheral artery stenosis |
| Potentially leading to amputation | 10072564 | Peripheral artery thrombosis |
| Potentially leading to amputation | 10074396 | Penetrating atherosclerotic ulcer |
| Potentially leading to amputation | 10075118 | Subperiosteal abscess |
| Potentially leading to amputation | 10075714 | Vasculitic ulcer |
| Potentially leading to amputation | 10076246 | Spontaneous amputation |

#### Appendix D Potentially clinically significant abnormalities criteria

# CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES for Phase 2/3 studies (oncology excepted) (From BTD-009536 May 21, 2014)

**Parameter PCSA** Comments **Clinical Chemistry** ALT By distribution analysis: Enzymes activities must be expressed in ULN, not in IU/L. >3 ULN Concept paper on DILI - FDA draft >5 ULN Guidance Oct 2007. >10 ULN Internal DILI WG Oct 2008. >20 ULN Categories are cumulative. First row is mandatory. Rows following one mentioning zero can be deleted. AST By distribution analysis: Enzymes activities must be expressed in ULN, not in IU/L. >3 ULN Concept paper on DILI - FDA draft >5 ULN Guidance Oct 2007. >10 ULN Internal DILI WG Oct 2008. >20 ULN Categories are cumulative. First row is mandatory. Rows following one mentioning zero can be deleted. Alkaline Phosphatase >1.5 ULN Enzymes activities must be expressed in ULN, not in IU/L. Concept paper on DILI - FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. Total Bilirubin >1.5 ULN Must be expressed in ULN, not in µmol/L or mg/L. Categories are cumulative. >2 ULN Concept paper on DILI - FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. >35% Total Bilirubin and TBILI>1.5 ULN Conjugated Bilirubin Conjugated bilirubin dosed on a case-by-case basis. ALT and Total Bilirubin ALT>3 ULN and TBILI>2 ULN Concept paper on DILI - FDA draft Guidance Oct 2007. Internal DILI WG Oct 2008. To be counted within a same treatment phase, whatever the interval between measurement.

#### CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

#### for Phase 2/3 studies (oncology excepted)

(From BTD-009536 May 21, 2014)

| Parameter | PCSA | | Comments |
|---|---|---|---|
| CPK | >3 ULN<br>>10 ULN | | FDA Feb 2005. Am J Cardiol April 2006. Categories are cumulative. First row is mandatory. Rows following one mentioning zero can be deleted. |
| CLcr (mL/min) (Estimated creatinine clearance based on the Cockcroft-Gault equation) | <15 (end stage renal disease) ≥15 - <30 (severe decrease in GFR) ≥30 - <60 (moderate decrease in GFR) ≥60 - <90 (mild decrease in GFR) ≥ 90 (normal GFR) | FDA draft Guidance<br>Pharmacokinetics i<br>impaired renal func<br>analysis, and impac<br>labeling | e 2010<br>n patients with<br>tion-study design, data |
| eGFR<br>(mL/min/1.73m2)<br>(Estimate of GFR<br>based on an<br>MDRD equation) | <15 (end stage renal disease) ≥15 - <30 (severe decrease in GFR) ≥30 - <60 (moderate decrease in GFR) ≥60 - <90 (mild decrease in GFR) ≥ 90 (normal GFR) | FDA draft Guidance<br>Pharmacokinetics i<br>impaired renal func<br>analysis, and impac<br>labeling | n patients with<br>tion-study design, data |
| Creatinine | • | (Adults)<br>le from baseline<br>lge from baseline | Benichou C., 1994. |
| Uric Acid<br>Hyperuricemia<br>Hypouricemia | >408 µmol/L<br><120 µmol/L | | Harrison- Principles of internal Medicine 17 <sup>th</sup> Ed., 2008. |
| Blood Urea Nitroger | n ≥17 mmol/L | | |
| Chloride | <80 mmol/L<br>>115 mmol/L | _ | |
| Sodium | ≤129 mmol/l<br>≥160 mmol/l | | |
| Potassium | <3 mmol/L<br>≥5.5 mmol/L | | FDA Feb 2005. |
| Total Cholesterol | ≥7.74 mmol/ | L | Threshold for therapeutic intervention. |
| Triglycerides | ≥4.6 mmol/L | | Threshold for therapeutic intervention. |
| Lipasemia | ≥3 ULN | | |
| Amylasemia | ≥3 ULN | | |

#### CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

#### for Phase 2/3 studies (oncology excepted)

(From BTD-009536 May 21, 2014)

| Parameter PCSA | | Comments |
|---|---|---|
| Glucose | | |
| Hypoglycaemia | ≤3.9 mmol/L and <lln< td=""><td>ADA May 2005.</td></lln<> | ADA May 2005. |
| Hyperglycaemia | ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) | ADA Jan 2008. |
| HbA1c | >8% | |
| Albumin | ≤25 g/L | |
| CRP | >2 ULN or >10 mg/L (if ULN not provided) | FDA Sept 2005. |
| Hematology | | |
| WBC | <3.0 Giga/L (Non-Black); <2.0 Giga/L | Increase in WBC: not relevant. |
| | (Black)<br>≥16.0 Giga/L | To be interpreted only if no differential count available. |
| Lymphocytes | >4.0 Giga/L | |
| Neutrophils | <1.5 Giga/L (Non-Black);<1.0 Giga/L (Black) | International Consensus meeting on drug-<br>induced blood cytopenias, 1991. |
| | | FDA criteria. |
| Monocytes | >0.7 Giga/L | |
| Basophils | >0.1 Giga/L | |
| Eosinophils | >0.5 Giga/L or >ULN (if ULN≥0.5 Giga/L) | Harrison- Principles of internal Medicine 17 <sup>th</sup> Ed., 2008. |
| Hemoglobin | ≤115 g/L (Male); ≤95 g/L (Female)<br>≥185 g/L (Male); ≥165 g/L (Female) | Criteria based upon decrease from baseline are more relevant than based on absolute value. Other categories for |
| | Decrease from Baseline ≥20 g/L | decrease from baseline can be used ( $\geq$ 30 g/L, $\geq$ 40 g/L, $\geq$ 50 g/L). |
| Hematocrit | ≤0.37 v/v (Male) ; ≤0.32 v/v (Female) | |
| | ≥0.55 v/v (Male) ; ≥0.5 v/v (Female) | |
| RBC | ≥6 Tera/L | Unless specifically required for particular drug development, the analysis is redundant with that of Hb. |
| | | Otherwise, consider FDA criteria. |
| Platelets | <100 Giga/L | International Consensus meeting on |
| | ≥700 Giga/L | drug-induced blood cytopenias, 1991. |


#### CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

#### for Phase 2/3 studies (oncology excepted)

(From BTD-009536 May 21, 2014)

| Parameter | PCSA | Comments |
|---|---|---|
| Urinalysis | | |
| pH | ≤4.6 | |
| | ≥8 | |
| Vital signs | | |
| HR | ≤50 bpm and decrease from baseline ≥20 bpm | To be applied for all positions (including missing) except STANDING. |
| | ≥120 bpm and increase from baseline≥20 bpm | |
| SBP | ≤95 mmHg and decrease from baseline ≥20mmHg | To be applied for all positions (including missing) except STANDING. |
| | ≥160 mmHg and increase from baseline<br>≥20 mmHg | |
| DBP | ≤45 mmHg and decrease from baseline ≥10 mmHg | To be applied for all positions (including missing) except STANDING. |
| | ≥110 mmHg and increase from baseline<br>≥10 mmHg | |
| Orthostatic Hypotension | | |
| Orthostatic SDB | | |
| Orthostatic DBP | ≤-20 mmHg<br>≤-10 mmHg | |
| Weight | ≥5% increase from baseline ≥5% decrease from baseline | FDA Feb 2007. |

#### CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

#### for Phase 2/3 studies (oncology excepted)

(From BTD-009536 May 21, 2014)

| Parameter | PCSA | Comments |
|---|---|---|
| ECG | | Ref.: ICH E14 guidance (2005) and E14 Q&A (2012), and Cardiac Safety Research Consortium White Paper on PR and QRS (Nada et al. Am Heart J. 2013; 165(4): 489-500) |
| HR | <50 bpm <50 bpm and decrease from baseline ≥20 bpm <40 bpm <40 bpm and decrease from baseline ≥20 bpm <30 bpm | Categories are cumulative |
| | <30 bpm and decrease from baseline ≥20 bpm >90 bpm >90 bpm and increase from baseline ≥20bpm >100 bpm >100 bpm and increase from baseline ≥20bpm >120 bpm >120 bpm >120 bpm >120 bpm and increase from baseline ≥20 bpm | Categories are cumulative |
| PR | >200 ms >200 ms and increase from baseline ≥25% >220 ms >220 ms >220 ms and increase from baseline ≥25% >240 ms >240 ms >240 ms and increase from baseline ≥25% | Categories are cumulative |
| QRS | >110 ms >110 msec and increase from baseline ≥25% >120 ms >120 ms and increase from baseline ≥25% | Categories are cumulative |


#### CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

#### for Phase 2/3 studies (oncology excepted)

(From BTD-009536 May 21, 2014)

| Parameter | PCSA | Comments |
|---|---|---|
| QT | >500 ms | |
| QTc | Absolute values (ms) | To be applied to any kind of QT correction formula. |
| | >450 ms | Absolute values categories are cumulative |
| | >480 ms | |
| | >500 ms | QTc >480 ms and ∆QTc>60 ms are the 2 PCSA categories to be identified in |
| | Increase from baseline | individual patients listings. |
| | Increase from baseline ]30-60] ms | |
| | Increase from baseline >60 ms | |

#### Appendix E Summary of statistical analyses

#### **EFFICACY ANALYSIS**

| Endpoint | Analysis population | Primary<br>analysis | Supportive analysis | Subgroup<br>analysis | Other analyses |
|---|---|---|---|---|---|
| Primary endpoint | | | | | |
| HbA1c: Change from baseline at Week 26, (sotagliflozin versus placebo) | ITT | ANCOVA (with missing values imputed by the retrieved dropouts or washout imputation method under MNAR framework): treatment, randomization stratum (HbA1c /metformin use/SBP at screening), and country as fixed effects, and baseline HbA1c value as a covariate | Tipping point analysis; | Subgroups: race, ethnicity, age, gender, baseline BMI, baseline HbA1c, baseline SBP, metformin use at screening, baseline eGFR, Duration of diabetes, and country | Summary statistics for observed values and changes from baseline by visit. Graphical presentations for mean changes from baseline (±SE) and mean values (±SE) by visit. By-visit summary and graph excluding measurements after rescue therapy. |
| Secondary endpoints | | | | | |
| HbA1c(sotagliflozin versus empagliflozin); 2-hour PPG reduction, body weight (sotagliflozin versus placebo only): Change from baseline to Week 26; SBP (for patients with baseline SBP ≥130 mmHg): Change from baseline to Week 12; SBP any baseline (sotagliflozin versus empagliflozin only): Change from baseline to Week 12 | ITT | ANCOVA (with missing values imputed by the retrieved dropouts or washout imputation method under MNAR framework): treatment, randomization stratum (HbA1c /metformin use /SBP at screening), and country as fixed effects, and baseline value as a covariate | Tipping point<br>analysis and<br>Completer<br>analysis for<br>HbA1c<br>(sotagliflozin<br>versus<br>empagliflozin) | For HbA1c<br>(sotagliflozin versus<br>empagliflozin):<br>similar to primary<br>endpoint subgroups | Summary statistics for observed values and changes from baseline by visit. Graphical presentations for mean changes from baseline (±SE) and mean values (±SE) by visit. SBP will be summarized descriptively at each visit for those with baseline SBP ≥140 mmHg |

## Version:3

Lexicon Pharmaceuticals Protocol No. EFC14867

| Endpoint | Analysis population | Primary<br>analysis | Supportive analysis | Subgroup<br>analysis | Other analyses |
|---|---|---|---|---|---|
| Other endpoints | | | | | |
| SBP (for patients with baseline SBP <130 mmHg), DBP, Serum creatinine, eGFR, UGE, UGCR, UACR, hemodynamic markers: change from Baseline | ITT | Summary statistics for observed values and changes from baseline by visit. In addition for UGE and UGCR, ANCOVA (with missing values imputed by the retrieved dropouts or washout imputation method under MNAR framework): treatment, randomization stratum (HbA1c /metformin use /SBP at screening), and country as fixed effects, and baseline value as a covariate | No | No | Graphical presentations for mean changes from baseline (±SE) and mean values (±SE) by visit as appropriate. |

Date of Issue: 15-Nov-2019

Covance Study ID: 000000155204

## Version:3 Lexicon Pharmaceuticals Protocol No. EFC14867

| Endpoint | Analysis population | Primary<br>analysis | Supportive analysis | Subgroup<br>analysis | Other analyses |
|---|---|---|---|---|---|
| Proportion of patients with HbA1c <6.5%, <7.0% at Week 26 | ITT | CMH method stratified on randomization strata (HbA1c /metformin use/SBP at screening), | CMH method stratified on randomization strata (HbA1c /metformin use/ SBP at: excluding patients with baseline HbA1c values <6.5% (for <6.5% responders) or <7% (for <7% responders) respectively | No | By-visit summary and graphs of HbA $_{1c}$ responders (<6.5%, <7%). By-visit frequency summary and graphs of HbA $_{1c}$ responders (<6.5%, <7%) excluding patients with baseline HbA $_{1c}$ values <6.5% or <7% respectively. |
| Proportion of patients, with reduction in body weight by ≥2%, ≥5%, and ≥10% from Baseline | ITT | By-visit frequency summary | No | No | By-visit graphical presentation as appropriate |
| Proportion of patients requiring rescue for hyperglycemia | ITT | Summary statistics | No | No | KM plot; List of patients rescued |

Date of Issue: 15-Nov-2019

Covance Study ID: 000000155204

## Version:3 Lexicon Pharmaceuticals Protocol No. EFC14867

| Endpoint | Analysis population | Primary<br>analysis | Supportive analysis | Subgroup<br>analysis | Other<br>analyses |
|---|---|---|---|---|---|
| ABPM Substudy | | | | | |
| Changes from Baseline to Week 12 and Week 26 in: | ABPM population | Summary statistics for observed values and | No | No | |
| Average 24-hour SBP and DBP, average adjusted awake time BP as measured by SBP and DBP with adjustment based on actigraphy, average adjusted awake time BP as measured by SBP and DBP with adjustment based on actigraphy for all patients participating substudy, patients with baseline average 24-hour SBP≥130 mmHg and patients with baseline average 24-hour SBP<130 mmHg. | | changes from baseline by visit. | | | |

Date of Issue: 15-Nov-2019

Covance Study ID: 000000155204

#### SAFETY ANALYSES

| Endpoint | Analysis<br>Population | Primary<br>analysis | Supportive<br>Analysis | Subgroup<br>analysis | Other analyses |
|---|---|---|---|---|---|
| Hypoglycemia | Safety | Follow safety guidelines Number (%) of patients with any hypoglycemia, severe hypoglycemia, documented symptomatic hypoglycemia during TEAE period, and incidence rates in 100 patient-years. | | Severe hypoglycemia or<br>documented symptomatic<br>hypoglycemia by subgroups: race,<br>age, gender, metformin use | KM plot time to first event of severe hypoglycemia or documented symptomatic hypoglycemia Documented symptomatic hypoglycemia maybe presented by <3.0 mmol/L (<54 mg/dL) as appropriate. |
| Adverse Events | Safety | Follow safety guidelines | No | Common TEAEs by subgroups: race, age, gender, baseline SBP, metformin use, baseline eGFR | |
| Clinical laboratory data | Safety | Follow safety guidelines | Descriptive | No | No |
| Vital signs | Safety | Follow safety guidelines | Descriptive | No | No |
| ECG, Physical examination | Safety | Follow safety guidelines | Frequency summary | No | No |

### Appendix F Study Flow Chart

| | Scre | ening Pe | riod | | | Doub | le-blind Tre | eatment P | eriod <sup>a</sup> | | | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screenin<br>g | Run-in | | | | | | | | | | |
| Visit | 1 | 2 | 3A<br>ABPM | 3<br>Rando-<br>mization | 4 | 5 | 6A<br>ABPM | 6 | 7 | 8A<br>ABPM | 8 | 9 |
| Week | Up to -4 | -2 | -1 | 0<br>Baseline | 4 | 8 | 12 | 12 | 18 | 26 | 26 | 30 |
| Day (window [days]) | | -14<br>(±3) | -7 | 1 | 28<br>(±3) | 56<br>(±3) | 83<br>(±3) | 84<br>(±3) | 126<br>(±5) | 181<br>(±5) | 182<br>(±5) | 210<br>(±5) |
| Informed consent | Х | | | | | | | | | | | |
| Interactive Response<br>Technology (IRT) contact | Х | Х | | Х | Х | Х | | Х | Х | | Х | Х |
| Inclusion criteria | Х | | | | | | | | | | | |
| Exclusion criteria | Х | | | Х | | | | | | | | |
| Demographics | Х | | | | | | | | | | | |
| Medical and surgical history | Х | | | | | | | | | | | |
| Medication history | Х | | | | | | | | | | | |
| Concomitant medication | X | Χ | | Х | Χ | Х | | Χ | Х | | Х | Х |
| Body weight, height <sup>c</sup> | Х | Χ | | Χ | Χ | Х | | Χ | Х | | Х | Х |
| Vital signs <sup>d</sup> | Х | Х | | Х | Х | Х | | Х | Х | | Х | Х |
| Physical examination: | | | | | | | | | | | | |
| Complete | Х | | | | | | | | | | Х | |
| Abbreviated <sup>e</sup> | | Х | | Х | Х | Х | | Х | Х | | | Х |
| Diet and exercise instruction | | Х | | Х | | | | | | | Х | |

| | Scre | ening Pe | riod | | | Doub | le-blind Tr | eatment P | erioda | | | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screenin<br>g | Ru | n-in | | | | | | | | | up <sup>b</sup> |
| Visit | 1 | 2 | 3A<br>ABPM | 3<br>Rando-<br>mization | 4 | 5 | 6A<br>ABPM | 6 | 7 | 8A<br>ABPM | 8 | 9 |
| Week | Up to -4 | -2 | -1 | 0<br>Baseline | 4 | 8 | 12 | 12 | 18 | 26 | 26 | 30 |
| Day (window [days]) | | -14<br>(±3) | -7 | 1 | 28<br>(±3) | 56<br>(±3) | 83<br>(±3) | 84<br>(±3) | 126<br>(±5) | 181<br>(±5) | 182<br>(±5) | 210<br>(±5) |
| Instruction on basic genitourinary (GU) hygiene and hydration | | Х | | Х | Х | Х | | Х | Х | | Х | |
| Randomization | | | | Х | | | | | | | | |
| Dispense glucose meter | | Х | | | | | | | | | | |
| Collect glucose meter | | | | | | | | | | | | Х |
| Dispense diary | | Х | | Х | Х | Х | | Х | Х | | Х | |
| Collect/review diary | | | | Х | Χ | Х | | Х | Х | | Х | Х |
| Instruction on diabetic ketoacidosis symptoms and glucose testing | | Х | | Х | Х | Х | | Х | Х | | Х | |
| Dispense investigational medicinal product (IMP) | | Х | | Х | Х | Х | | Х | Х | | | |
| IMP accounting and compliance | | | | Х | Χ | Х | | Х | Х | | Х | |
| SMBG <sup>f</sup> | | Х | | Х | Х | Х | | Х | Х | | Х | |
| 12-lead electrocardiogram <sup>g</sup> | | Χ | | | | | | | | | Х | |
| MMTT/Postprandial glucose <sup>h</sup> | | | | Х | | | | | | | Х | |

| | Scre | ening Pe | riod | | | Doub | ole-blind Tr | eatment P | eriod <sup>a</sup> | | | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screenin<br>g | Ru | ın-in | | | | | | | | | up <sup>b</sup> |
| Visit | 1 | 2 | 3A<br>ABPM | 3<br>Rando-<br>mization | 4 | 5 | 6A<br>ABPM | 6 | 7 | 8A<br>ABPM | 8 | 9 |
| Week | Up to -4 | -2 | -1 | 0<br>Baseline | 4 | 8 | 12 | 12 | 18 | 26 | 26 | 30 |
| Day (window [days]) | | -14<br>(±3) | -7 | 1 | 28<br>(±3) | 56<br>(±3) | 83<br>(±3) | 84<br>(±3) | 126<br>(±5) | 181<br>(±5) | 182<br>(±5) | 210<br>(±5) |
| Ambulatory blood pressure monitoring (ABPM) <sup><i>i</i></sup> | | | Х | | | | Х | | | Х | | |
| Central Laboratory testing <sup>j</sup> | | | | | | | | | | | | |
| Fasting plasma glucose (FPG) <sup>k</sup> | Х | | | Х | Х | Х | | Х | Х | | Х | |
| HbA1c | Х | | | Х | | Х | | Х | | | Х | |
| Chemistry | Х | | | Х | Χ | | | Х | | | Х | Х |
| Hematology | Х | | | Х | Χ | | | Х | | | Х | |
| Fasting lipids | | | | Х | | | | | | | Х | |
| Pregnancy test (WOCBP) | Х | | | Х | Χ | Х | | Χ | Х | | Х | |
| FSH and/or estradiol as needed <sup>/</sup> | Х | | | | | | | | | | | |
| Sotagliflozin plasma concentration <sup>m</sup> | | | | | Х | | | | Х | | Х | |
| Hemodynamic markers <sup>n</sup> | | | | Х | | | | Х | | | Х | |
| Urinalysis with microscopy <sup>o</sup> | Х | | | Х | | | | | | | Х | |

| | Scre | ening Per | riod | | | Doub | le-blind Tr | eatment P | eriod <sup>a</sup> | | | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screenin<br>g | Run-in | | | | | | | | | | |
| Visit | 1 | 2 | 3A<br>ABPM | 3<br>Rando-<br>mization | 4 | 5 | 6A<br>ABPM | 6 | 7 | 8A<br>ABPM | 8 | 9 |
| Week | Up to -4 | -2 | -1 | 0<br>Baseline | 4 | 8 | 12 | 12 | 18 | 26 | 26 | 30 |
| Day (window [days]) | | -14<br>(±3) | -7 | 1 | 28<br>(±3) | 56<br>(±3) | 83<br>(±3) | 84<br>(±3) | 126<br>(±5) | 181<br>(±5) | 182<br>(±5) | 210<br>(±5) |
| Collection of home overnight urine for albumin, total protein, creatinine, calcium, phosphorus, magnesium, and glucosep <sup>p</sup> | | | | Х | | | | Х | | | Х | |
| Urine NMP-22 and cytologyq <sup>q</sup> | | | | | To be | assessed as | clinically indic | ated | | | | |
| Evaluate for glycemic rescue | | | | | To b | e assessed | and reported t | hroughout th | e treatment p | period | | |
| Hypoglycemia | | | | T | To be assess | ed and repo | rted throughou | ut the study <sup>t</sup> | | | | |
| AEs/SAEs/AESI/EOSI | | | | 7 | o be assess | ed and repo | rted throughou | ut the study <sup>t</sup> | | | | |

a If a patient discontinues treatment with IMP early during the Double-blind Treatment Period, the patient will have a Premature EOT Visit (similar to Visit 8) and a Follow-up Visit 4 weeks ± 5 days after the last dose of IMP. In addition, every effort will be made to have the patient return to the site at the time corresponding to their scheduled visits, particularly the Week 26 Visit. If the patient does not agree to a site visit, they will be contacted by telephone to inquire about safety status.

- b The Follow-up Visit will take place 4 weeks ± 5 days after the last dose of IMP. All attempts will be made to contact the patient to inquire about safety status.
- c Height will be measured only at Screening Visit.
- d Vital sign measurements (sitting BP and heart rate): At the Screening Visit, BP will be measured on both arms to identify and select the appropriate arm for future measurements. Three separate seated BP and heart rate measurements should be taken with at least 1 minute between readings, following a 5-minute rest period and prior to phlebotomy. Assessment for volume contraction and correct volume status, if indicated, will be done before randomization.
- e The abbreviated physical examination should focus on cardiac and respiratory systems, as well as any areas important for assessment of adverse events if necessary.

#### Version:3

Lexicon Pharmaceuticals Protocol No. EFC14867

**Date of Issue: 15-Nov-2019**Covance Study ID: 000000155204

- f The SMBG is to be performed fasting (before first meal of the day) for at least 3 days in the week prior to each study visit. The SMBG should be performed in case of hypoglycemia symptoms; any SMBG values ≤70 mg/dL (≤3.9 mmol/L) should be documented in the diary and collected in the hypoglycemia event CRF. The SMBG will be presented as equivalent SMPG.
- g The 12-lead ECG should be performed after the patient has spent at least 10 minutes in supine position and prior to IMP administration. The ECG results will be evaluated as "normal" or "abnormal".
- h Plasma postprandial glucose will be assessed at Baseline Week 0 and Week 26, 2 hours after consuming a standard mixed liquid breakfast meal via an MMTT.
- i Visit for ABPM for a subset of patients (180 patients) will occur 1 week before the Randomization Visit; patients will return the ABPM device by mail after 24-hour monitoring is complete. Patients will also have additional in-person visits for placement of the ABPM device on the day before Week 12 and 26 visits. At least 70% recording of the expected BP recording is needed in each 24-hour period. The measurement will be done on the nondominant upper arm. Patients who discontinue the IMP before the visit for ABPM will not continue in the ABPM substudy post-IMP discontinuation. Patients who receive rescue therapy but remain on IMP will continue on the ABPM substudy as planned.
- j With the exception of PPG, all laboratory assessments will occur prior to IMP administration on the day of the visit. All visit dates will be scheduled based on the date of randomization with a ±3-day visit window allowed during the core treatment period, except for Visits 7, 8A, 8, and 9, when a ±5 days visit window will apply.
- k The FPG collection will be performed on the morning of visit.
- I Serum pregnancy testing will be performed only at Screening and urine pregnancy testing is performed at subsequent visits. Serum pregnancy test results must be reviewed prior to the Run-in Phase for all women of childbearing potential. Any positive urine test results must be confirmed based on serum pregnancy test. The Investigator may perform additional tests at their discretion or as required by local regulations. For women of non-productive potentials, follicle-stimulating hormone [FSH] and/or estradiol levels should be tested in case the definition of postmenopausal or premenopausal can't be satisfied, eg, no medical document of hysterectomy or cessation of menses without an alternative medical cause is <12 months.
- m Plasma concentration samples (ie, of sotagliflozin and sotaglifl
- n Hemodynamic markers including PRA, aldosterone, angiotensinogen 1, angiotensinogen 2, and glucagon will be checked to provide better characterization of hemodynamic markers in relation to sotagliflozin treatment.
- o Urinalysis will include urine dipstick and microscopy. Dipstick will include assessment of specific gravity, pH, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase. Microscopy will include, but not be limited to, detection of formed cellular elements, casts, bacteria, yeast, parasites, and crystals in centrifuged urine sediment. In the event of abnormal urinalysis findings suspicious of UTI, urine culture should be performed. Positive urine culture determination will be based upon the criteria of the reporting laboratory. Additionally, urine culture should be performed if at any point the Investigator suspects the presence of a UTI.
- p Patients will collect overnight urine on Week 0, 12, and 26 (Visits 3, 6 and 8). In the night prior to the visits, the urine before sleep will be discarded and the urine during sleep and the first morning urine (after getting up) will be collected. The visits should be rescheduled to allow for urine collection in case a patient missed it. Urinary albumin, total protein, creatinine, calcium (adjusted for creatinine), phosphorus (adjusted for serum phosphorus and creatinine), magnesium (adjusted for serum magnesium and urinary creatinine), and glucose will be assessed.
- q Urine NMP-22 and cytology should only be performed when clinically indicated in cases of unexplained hematuria, and should be assessed by the central laboratory.

All SAEs, AESI, and EOSI will be collected starting from signing informed consent and continue until the end of the study (Note: For patients who discontinue treatment >2 weeks before Week 26, safety data will be collected until scheduled study end). All AEs that occur during treatment should be followed until study completion (or until patients leave the study) or until the event has resolved, the condition has stabilized or the patient is lost to follow-up, whichever comes earlier. All patients will have a Follow-up visit 4 weeks ± 5 days after the last dose of IMP to collect safety information.